CLINICAL TRIAL: NCT02055976
Title: A Phase 2 Double Blind, Parallel Group, Placebo Controlled, Randomized, Dose Ranging Study To Assess The Efficacy, Safety And Tolerability Of Pf-04950615 Following Twice Monthly Subcutaneous Doses In Hypercholesterolemic Japanese Subjects Who Are Receiving A Stable Dose Of Atorvastatin Or Treatment Naïve.
Brief Title: Dose Ranging Study Of Bococizumab (PF-04950615; RN316) In Hypercholesterolemic Japanese Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B1481036
Record Dates: First submitted 2014-01-22; First posted 2014-02-05 (Estimated); Results first posted 2019-02-08 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2018-09

CONDITIONS: Hypercholesterolemia
Keywords: PF-04950615; Japan
MeSH Terms: conditions — Hypercholesterolemia | interventions — bococizumab; Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Population A (Experimental): A total of 9 groups in two population. Population A comprises hypercholesterolemic Japanese subjects whose LDL-C is not controlled by a stable dose of atorvastatin. A subject who is receiving a stable dose of atorvastatin will be randomized into one out of 5 dose groups.
  Interventions: Drug: Bococizumab (PF-04950615;RN316); Drug: Placebo; Drug: Ezetimibe
- Population B (Experimental): A total of 9 groups in two population. Population B comprises hypercholesterolemic Japanese subjects who are naïve for a treatment by lipid lowering drug and whose fasting LDL-cholesterol is not controlled. A subject who is treatment naïve will be randomized into one out of 4 dose groups.
  Interventions: Drug: Bococizumab (PF-04950615;RN316); Drug: Placebo

INTERVENTIONS:
Drug: Bococizumab (PF-04950615;RN316) — Atorvastatin plus PF-04950615 50 mg subcutaneous administration at every two weeks (Q14D SC) for 16 week
  Arms: Population A
Drug: Bococizumab (PF-04950615;RN316) — Atorvastatin plus PF-04950615 100 mg Q14D SC for 16 week
  Arms: Population A
Drug: Bococizumab (PF-04950615;RN316) — Atorvastatin plus PF-04950615 150 mg Q14D SC for 16 week
  Arms: Population A
Drug: Placebo — Atorvastatin plus PF-04950615 Placebo Q14D SC for 16 week
  Arms: Population A
Drug: Ezetimibe — Atorvastatin plus Ezetimibe 10 mg oral administration once daily for 16 week (open)
  Arms: Population A
Drug: Bococizumab (PF-04950615;RN316) — 50 mg Q14D SC for 16 week
  Arms: Population B
Drug: Bococizumab (PF-04950615;RN316) — 100 mg Q14D SC for 16 week
  Arms: Population B
Drug: Bococizumab (PF-04950615;RN316) — 150 mg Q14D SC for 16 week
  Arms: Population B
Drug: Placebo — Placebo Q14D SC for 16 week
  Arms: Population B

SUMMARY:
The purpose of this study is to evaluate the low density lipoprotein cholesterol (LDL-C) lowering effect of Bococizumab (PF-04950615;RN316) administered subcutaneously at every two weeks (Q14D) in hypercholesterolemic Japanese subjects whose LDL-C is not controlled by a stable dose of atorvastatin, or who are naïve to a treatment by lipid lowering drug and whose LDL-C is not controlled.

ELIGIBILITY:
Inclusion Criteria:

* Subjects whose LDL-C is not controlled by a stable dose of atorvastatin (Population A).
* Subjects who are naïve to a treatment by lipid lowering drug and whose LDL-C is not controlled (Population B).

Exclusion Criteria:

* Severe acute or chronic medical or psychiatric condition or laboratory abnormality.
* Pregnant females; breastfeeding females; males and females of childbearing potential; males and females of childbearing potential who are unwilling or unable to use a highly effective method of contraception.
* Subjects who were administered or prior exposed to PF-04950615 and/or anti-body targeting PCSK9.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- Japan (9):
  - Maebashi Hirosegawa Clinic, Maebashi, Gunma
  - Yokohama Minoru Clinic, Yokohama, Kanagawa
  - Heishinkai Medical Group Incorporated OCROM Clinic, Suita, Osaka
  - Meiwa Hospital, Chiyoda-ku, Tokyo
  - Tokyo-Eki Center-building Clinic, Chuo-ku, Tokyo
  - Heishinkai Medical Group Incorporated ToCROM Clinic, Shinjuku-ku, Tokyo
  - Clinical Research Hospital Tokyo, Shinjuku-ku, Tokyo
  - Oda Clinic, Shinjuku-ku, Tokyo
  - Sekino Hospital, Toshima-ku, Tokyo

REFERENCES:
- [Derived] Wang EQ, Kaila N, Plowchalk D, Gibiansky L, Yunis C, Sweeney K. Population PK/PD modeling of low-density lipoprotein cholesterol response in hypercholesterolemic participants following administration of bococizumab, a potent anti-PCSK9 monoclonal antibody. CPT Pharmacometrics Syst Pharmacol. 2023 Dec;12(12):2013-2026. doi: 10.1002/psp4.13050. Epub 2023 Nov 22. PMID 37994400
- [Derived] Yokote K, Suzuki A, Li Y, Matsuoka N, Teramoto T. Pharmacokinetics and exploratory efficacy biomarkers of bococizumab, an anti-PCSK9 monoclonal antibody, in hypercholesterolemic Japanese subjects . Int J Clin Pharmacol Ther. 2019 Dec;57(12):575-589. doi: 10.5414/CP203418. PMID 31549625
- [Derived] Yokote K, Kanada S, Matsuoka O, Sekino H, Imai K, Tabira J, Matsuoka N, Chaudhuri S, Teramoto T. Efficacy and Safety of Bococizumab (RN316/PF-04950615), a Monoclonal Antibody Against Proprotein Convertase Subtilisin/Kexin Type 9, in Hypercholesterolemic Japanese Subjects Receiving a Stable Dose of Atorvastatin or Treatment-Naive - Results From a Randomized, Placebo-Controlled, Dose-Ranging Study. Circ J. 2017 Sep 25;81(10):1496-1505. doi: 10.1253/circj.CJ-16-1310. Epub 2017 May 23. PMID 28539539
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1481036&StudyName=Dose%20Ranging%20Study%20Of%20PF-04950615%20In%20Hypercholesterolemic%20Japanese%20Subjects

RESULTS

PARTICIPANT FLOW:
Groups:
- Atorvastatin + PF-04950615 50 mg: Participants with fasting lipoprotein cholesterol (LDL-C) level (greater than or equal to [>=]100 milligram per deciliter [mg/dL]) received atorvastatin along with PF-04950615 50 milligram (mg) subcutaneous injection, once daily on Day 1, 15, 29, 43, 57, 71, 85 and 99. Participants were on self-administered stable background atorvastatin therapy.
- Atorvastatin + PF-04950615 100 mg: Participants with fasting LDL-C level (>=100 [mg/dL]) received atorvastatin along with PF-04950615 100 mg subcutaneous injection, once daily on Day 1, 15, 29, 43, 57, 71, 85 and 99. Participants were on self-administered stable background atorvastatin therapy.
- Atorvastatin + PF-04950615 150 mg: Participants with fasting LDL-C level (>=100 [mg/dL]) received atorvastatin along with PF-04950615 150 mg subcutaneous injection, once daily on Day 1, 15, 29, 43, 57, 71, 85 and 99. Participants were on self-administered stable background atorvastatin therapy.
- Atorvastatin + PF-04950615 Placebo: Participants with fasting LDL-C level (>=100 [mg/dL]) received atorvastatin along with PF-04950615 placebo subcutaneous injection, once daily on Day 1, 15, 29, 43, 57, 71, 85 and 99. Participants were on self-administered stable background atorvastatin therapy.
- Atorvastatin + Ezetimibe 10 mg: Participants with fasting LDL-C level (>=100 [mg/dL]) received atorvastatin along with ezetimibe 10 mg tablet orally, once daily from Day 1 up to Day 112. Participants were on self-administered stable background atorvastatin therapy.
- PF-04950615 50 mg: Participants with fasting LDL-C level (>=130 [mg/dL]) received PF-04950615 50 mg, subcutaneous injection, once daily on Day 1, 15, 29, 43, 57, 71, 85 and 99. Participants were naive to a treatment by lipid lowering drug.
- PF-04950615 100 mg: Participants with fasting LDL-C level (>=130 [mg/dL]) received PF-04950615 100 mg, subcutaneous injection, once daily on Day 1, 15, 29, 43, 57, 71, 85 and 99. Participants were naive to a treatment by lipid lowering drug.
- PF-04950615 150 mg: Participants with fasting LDL-C level (>=130 [mg/dL]) received PF-04950615 150 mg, subcutaneous injection, once daily on Day 1, 15, 29, 43, 57, 71, 85 and 99. Participants were naive to a treatment by lipid lowering drug.
- PF-04950615 Placebo: Participants with fasting LDL-C level (>=130 [mg/dL]) received PF-04950615 placebo, subcutaneous injection, once daily on Day 1, 15, 29, 43, 57, 71, 85 and 99. Participants were naive to a treatment by lipid lowering drug.
Period: Overall Study
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Started | 25 | 24 | 24 | 26 | 22 | 25 | 25 | 24 | 23
Completed | 25 | 24 | 23 | 25 | 22 | 24 | 23 | 24 | 23
Not Completed | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Does not meet entrance criteria | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all randomized and non-randomized participants who were administered at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo | Total
Number analyzed (Participants) | 25 | 24 | 24 | 26 | 22 | 25 | 25 | 24 | 23 | 218
Age, Customized [Count of Participants; unit: Participants]
  Less than (<) 18 years | 0 (8.9) | 0 (12.2) | 0 (8.6) | 0 (11.2) | 0 (10.7) | 0 (8.4) | 0 (10.6) | 0 (8.1) | 0 (11.7) | 0
  18-44 years | 1 | 3 | 1 | 3 | 2 | 1 | 3 | 3 | 2 | 19
  45-64 years | 18 | 10 | 16 | 14 | 14 | 16 | 14 | 20 | 12 | 134
  Greater than or equal to (>=) 65 years | 6 | 11 | 7 | 9 | 6 | 8 | 8 | 1 | 9 | 65
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 12 | 13 | 10 | 13 | 15 | 9 | 10 | 100
  Male | 17 | 14 | 12 | 13 | 12 | 12 | 10 | 15 | 13 | 118

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Fasting Low Density Lipoprotein-Cholesterol (LDL-C) at Day 85
Description: LDL-C is cholesterol in the bloodstream that is carried by low density lipoprotein. Fasting was required at least 10 hours before blood sample collection. Baseline was defined as the mean of the last two non-missing measurements collected prior to the first dose of study treatment. Both measurements must be within 10 days prior to the first dose of study treatment; if only one measurement was available 10 days prior to the first dose of study treatment, then that measurement served as the baseline value. Percent change from baseline = ([observed value divided by baseline value] minus 1) multiplied by 100.
Time Frame: Baseline, Day 85
Population: Full analysis set (FAS) included all the participants who were randomized and administered at least 1 dose of study treatment.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- PF-04950615 50 mg: Participants with fasting LDL-C level (>=130 [mg/dL]) received PF-04950615 50 mg, subcutaneous injection, once daily on Day 1, 15, 29, 43, 57, 71, 85 and 99. Participants were naïve to a treatment by lipid lowering drug.
- PF-04950615 100 mg: Participants with fasting LDL-C level (>=130 [mg/dL]) received PF-04950615 100 mg, subcutaneous injection, once daily on Day 1, 15, 29, 43, 57, 71, 85 and 99. Participants were naïve to a treatment by lipid lowering drug.
- PF-04950615 150 mg: Participants with fasting LDL-C level (>=130 [mg/dL]) received PF-04950615 150 mg, subcutaneous injection, once daily on Day 1, 15, 29, 43, 57, 71, 85 and 99. Participants were naïve to a treatment by lipid lowering drug.
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
percent change | -55.65 (15.748) [-60.388 to -49.639] | -68.25 (18.769) [-77.547 to -66.313] | -74.00 (13.848) [-82.354 to -71.066] | -5.91 (14.323) [-10.453 to 0.102] | -18.56 (15.968) | -47.25 (17.699) | -62.24 (16.097) | -65.89 (10.779) | -1.21 (14.815)
Statistical Analysis 1: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; Adjusted mean difference and 2-sided 95% confidence interval were derived from the mixed-effect model for repeated measures (MMRM) model with fixed effects for treatment, visit, baseline value, treatment by visit interaction, and baseline by visit interaction; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-value (adjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -49.838, 95% CI 2-sided [-57.335 to -42.340], Standard Error of Mean 3.775
Statistical Analysis 2: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; Adjusted mean difference and 2-sided 95% confidence interval were derived from the MMRM model with fixed effects for treatment, visit, baseline value, treatment by visit interaction, and baseline by visit interaction; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-value (adjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -66.754, 95% CI 2-sided [-74.523 to -58.986], Standard Error of Mean 3.912
Statistical Analysis 3: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (adjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -71.534, 95% CI 2-sided [-79.284 to -63.784], Standard Error of Mean 3.903
Statistical Analysis 4: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (adjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -47.531, 95% CI 2-sided [-55.511 to -39.551], Standard Error of Mean 4.016
Statistical Analysis 5: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (adjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -62.624, 95% CI 2-sided [-70.557 to -54.691], Standard Error of Mean 3.993
Statistical Analysis 6: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (adjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -64.268, 95% CI 2-sided [-72.128 to -56.409], Standard Error of Mean 3.955

2. Primary Outcome: Percent Change From Baseline in Fasting Low Density Lipoprotein-Cholesterol (LDL-C) at Day 113
Description: as for outcome 1
Time Frame: Baseline, Day 113
Population: FAS included all the participants who were randomized and administered at least 1 dose of study treatment. Here, number of participants analyzed (N) signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 23 | 23
percent change | -54.41 (12.062) [-60.388 to -49.639] | -64.46 (19.149) [-77.547 to -66.313] | -69.98 (19.074) [-82.354 to -71.066] | -12.10 (12.727) [-10.453 to 0.102] | -20.55 (18.682) | -44.94 (19.641) | -61.79 (15.476) | -66.98 (12.396) | 0.39 (16.246)
Statistical Analysis 1: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (adjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -42.293, 95% CI 2-sided [-49.417 to -35.168], Standard Error of Mean 3.587
Statistical Analysis 2: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (adjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -56.262, 95% CI 2-sided [-63.603 to -48.921], Standard Error of Mean 3.696
Statistical Analysis 3: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (adjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -61.384, 95% CI 2-sided [-68.733 to -54.035], Standard Error of Mean 3.700
Statistical Analysis 4: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (adjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -47.578, 95% CI 2-sided [-56.067 to -39.088], Standard Error of Mean 4.273
Statistical Analysis 5: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (adjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -63.346, 95% CI 2-sided [-71.776 to -54.915], Standard Error of Mean 4.244
Statistical Analysis 6: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (adjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -66.691, 95% CI 2-sided [-75.088 to -58.295], Standard Error of Mean 4.226

3. Secondary Outcome: Low Density Lipoprotein-Cholesterol (LDL-C)
Description: LDL-C is cholesterol in the bloodstream that is carried by low density lipoprotein. Fasting was required at least 10 hours before blood sample collection. Baseline was defined as the mean of the last two non-missing measurements collected prior to the first dose of study treatment. Both measurements must be within 10 days prior to the first dose of study treatment; if only one measurement was available 10 days prior to the first dose of study treatment, then that measurement served as the baseline value.
Time Frame: Baseline, Day 5, 8, 15, 22, 29, 36, 43, 50, 57, 71, 85, 99, 106, 113, 127, 141, 155, 169
Population: FAS included all the participants who were randomized and administered at least 1 dose of study treatment. Here, 'Number analyzed' = Participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 26 | 22 | 25 | 25 | 24 | 23
mg/dL
  Baseline | 135.36 (23.652) | 123.85 (20.585) | 129.19 (17.769) | 135.90 (24.697) | 135.36 (24.745) | 164.22 (25.839) | 158.00 (20.004) | 159.90 (19.800) | 155.22 (23.096)
  Day 5: number analyzed (Participants) | 25 | 23 | 23 | 26 | 22 | 25 | 25 | 24 | 22
  Day 5 | 86.72 (24.917) | 71.83 (26.020) | 76.04 (17.111) | 130.35 (22.280) | 111.50 (23.118) | 128.68 (30.905) | 120.20 (21.352) | 114.63 (30.177) | 165.09 (22.880)
  Day 8: number analyzed (Participants) | 25 | 24 | 24 | 25 | 21 | 25 | 24 | 22 | 23
  Day 8 | 70.36 (18.932) | 55.38 (28.309) | 57.71 (16.433) | 132.08 (21.244) | 105.86 (21.070) | 118.20 (33.823) | 102.63 (26.577) | 96.50 (36.130) | 167.22 (23.537)
  Day 15 | 73.76 (18.807) | 51.96 (23.921) | 39.00 (16.395) | 132.50 (19.449) | 102.64 (19.458) | 113.28 (36.371) | 80.44 (25.366) | 77.08 (25.943) | 165.39 (21.148)
  Day 22: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 22 | 49.08 (19.577) | 37.58 (20.011) | 31.00 (11.176) | 133.27 (19.359) | 101.68 (21.825) | 90.32 (34.956) | 67.29 (26.527) | 67.71 (32.399) | 166.04 (15.741)
  Day 29: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 25 | 25 | 24 | 22
  Day 29 | 61.56 (24.316) | 48.29 (21.814) | 34.26 (13.965) | 129.60 (23.381) | 107.50 (23.299) | 93.36 (36.718) | 65.20 (17.970) | 63.58 (23.404) | 168.14 (24.032)
  Day 36: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 36 | 44.40 (19.967) | 35.13 (17.306) | 29.52 (11.233) | 128.50 (23.930) | 103.05 (26.462) | 80.64 (34.744) | 60.67 (19.257) | 60.75 (27.619) | 154.00 (22.815)
  Day 43 | 58.24 (21.357) | 39.63 (20.342) | 31.83 (11.750) | 126.23 (14.356) | 104.95 (23.941) | 87.76 (36.555) | 64.84 (19.882) | 61.83 (29.732) | 167.30 (21.850)
  Day 50: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Day 50 | 39.76 (16.042) | 32.33 (16.578) | 29.96 (11.400) | 127.92 (20.392) | 106.23 (21.728) | 76.96 (32.194) | 57.91 (20.889) | 59.29 (28.406) | 158.83 (17.031)
  Day 57: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 57 | 56.88 (18.306) | 37.21 (18.352) | 29.61 (11.053) | 125.27 (20.330) | 99.27 (26.705) | 81.32 (33.628) | 63.54 (25.072) | 55.75 (26.272) | 152.91 (15.395)
  Day 71: number analyzed (Participants) | 24 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 71 | 61.50 (22.683) | 36.29 (18.196) | 33.13 (13.384) | 130.31 (21.031) | 109.18 (26.412) | 90.96 (34.188) | 60.63 (24.315) | 57.33 (25.237) | 156.70 (25.663)
  Day 85: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Day 85 | 58.96 (19.650) | 38.00 (19.077) | 33.91 (19.400) | 126.38 (21.478) | 110.64 (33.530) | 86.64 (30.447) | 59.83 (27.495) | 54.71 (18.388) | 151.30 (21.137)
  Day 99: number analyzed (Participants) | 25 | 24 | 22 | 25 | 22 | 25 | 24 | 24 | 23
  Day 99 | 66.48 (23.208) | 41.96 (18.995) | 38.09 (25.183) | 125.80 (15.992) | 106.14 (31.001) | 93.80 (29.672) | 61.67 (31.175) | 54.25 (20.339) | 163.70 (17.778)
  Day 106: number analyzed (Participants) | 25 | 24 | 22 | 25 | 22 | 25 | 23 | 24 | 23
  Day 106 | 45.16 (20.874) | 32.13 (18.059) | 37.36 (24.849) | 127.76 (17.973) | 104.14 (25.496) | 84.52 (29.679) | 57.00 (25.719) | 57.42 (22.654) | 155.57 (17.010)
  Day 113: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 23 | 23
  Day 113 | 62.17 (20.417) | 42.88 (19.427) | 38.48 (24.346) | 118.88 (22.883) | 107.32 (30.459) | 89.44 (29.798) | 61.48 (28.511) | 53.39 (20.954) | 153.30 (16.255)
  Day 127: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 25 | 23 | 24 | 23
  Day 127 | 108.16 (21.893) | 86.71 (27.414) | 61.87 (33.267) | 131.92 (21.922) | 132.73 (29.660) | 137.00 (36.894) | 87.22 (42.031) | 78.96 (25.696) | 161.17 (24.383)
  Day 141: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 24 | 23
  Day 141 | 126.13 (26.555) | 111.38 (24.588) | 95.30 (37.497) | 129.32 (20.860) | 139.14 (38.095) | 160.80 (37.487) | 130.22 (40.707) | 103.08 (34.759) | 163.52 (22.224)
  Day 155: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 23 | 23 | 24 | 23
  Day 155 | 126.52 (23.631) | 113.75 (19.236) | 110.57 (26.678) | 133.92 (23.240) | 139.45 (35.880) | 165.17 (31.251) | 140.78 (29.645) | 119.54 (32.896) | 158.17 (15.135)
  Day 169: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 24 | 23 | 23 | 22
  Day 169 | 131.28 (25.988) | 123.42 (25.782) | 124.04 (24.453) | 129.28 (24.576) | 140.91 (39.309) | 168.50 (28.657) | 154.52 (21.715) | 137.13 (32.817) | 168.55 (19.767)

4. Secondary Outcome: Change From Baseline in Low Density Lipoprotein-Cholesterol (LDL-C) at Day 85 and Day 113
Description: LDL-C is cholesterol in the bloodstream that is carried by low density lipoprotein. Fasting was required at least 10 hours before blood sample collection. Baseline was defined as the mean of the last two non-missing measurements collected prior to the first dose of study treatment. Both measurements must be within 10 days prior to the first dose of study treatment; if only one measurement was available 10 days prior to the first dose of study treatment, then that measurement served as the baseline value. Change from baseline = observed value minus baseline value.
Time Frame: Baseline, Day 85, 113
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 26 | 22 | 25 | 25 | 24 | 23
mg/dL
  Change at Day 85: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Change at Day 85 | -76.40 (26.447) | -85.85 (28.977) | -95.11 (21.145) | -9.52 (21.041) | -24.73 (23.125) | -77.58 (29.943) | -99.28 (32.550) | -105.19 (19.833) | -3.91 (23.632)
  Change at Day 113: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 23 | 23
  Change at Day 113 | -73.33 (18.047) | -80.98 (28.902) | -90.54 (28.496) | -17.48 (20.767) | -28.05 (23.663) | -74.78 (34.970) | -97.63 (25.545) | -107.57 (21.765) | -1.91 (20.147)
Statistical Analysis 1: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; Day 85 : Adjusted mean difference and 2-sided 95% confidence interval were derived from the MMRM model with fixed effects for treatment, visit, baseline value, treatment by visit interaction, and baseline by visit interaction; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -67.254, 95% CI 2-sided [-76.757 to -57.752], Standard Error of Mean 4.785
Statistical Analysis 2: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -87.122, 95% CI 2-sided [-96.969 to -77.275], Standard Error of Mean 4.959
Statistical Analysis 3: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -93.327, 95% CI 2-sided [-103.153 to -83.501], Standard Error of Mean 4.949
Statistical Analysis 4: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -71.724, 95% CI 2-sided [-84.128 to -59.321], Standard Error of Mean 6.243
Statistical Analysis 5: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -96.206, 95% CI 2-sided [-108.541 to -83.872], Standard Error of Mean 6.209
Statistical Analysis 6: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; Day 85: Adjusted mean difference and 2-sided 95% confidence interval were derived from the MMRM model with fixed effects for treatment, visit, baseline value, treatment by visit interaction, and baseline by visit interaction; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -98.533, 95% CI 2-sided [-110.743 to -86.323], Standard Error of Mean 6.145
Statistical Analysis 7: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; Day 113: Adjusted mean difference and 2-sided 95% confidence interval were derived from the MMRM model with fixed effects for treatment, visit, baseline value, treatment by visit interaction, and baseline by visit interaction; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -56.225, 95% CI 2-sided [-65.630 to -46.819], Standard Error of Mean 4.736
Statistical Analysis 8: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -73.813, 95% CI 2-sided [-83.507 to -64.119], Standard Error of Mean 4.881
Statistical Analysis 9: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -81.239, 95% CI 2-sided [-90.939 to -71.538], Standard Error of Mean 4.885
Statistical Analysis 10: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -72.573, 95% CI 2-sided [-84.461 to -60.684], Standard Error of Mean 5.983
Statistical Analysis 11: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -96.222, 95% CI 2-sided [-108.039 to -84.405], Standard Error of Mean 5.948
Statistical Analysis 12: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; Day 113:Adjusted mean difference and 2-sided 95% confidence interval were derived from the MMRM model with fixed effects for treatment, visit, baseline value, treatment by visit interaction, and baseline by visit interaction; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -102.184, 95% CI 2-sided [-113.945 to -90.424], Standard Error of Mean 5.919

5. Secondary Outcome: Total Cholesterol (TC)
Description: Total cholesterol is the sum of all the cholesterol within the blood. Fasting was required at least 10 hours before blood sample collection. Baseline was defined as the mean of the last two non-missing measurements collected prior to the first dose of study treatment. Both measurements must be within 10 days prior to the first dose of study treatment; if only one measurement was available 10 days prior to the first dose of study treatment, then that measurement served as the baseline value.
Time Frame: Baseline, Day 5, 8, 15, 22, 29, 36, 43, 50, 57, 71, 85, 99, 106, 113, 127, 141, 155, 169
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 26 | 22 | 25 | 25 | 24 | 23
mg/dL
  Baseline | 214.16 (30.658) | 210.29 (21.594) | 211.71 (23.065) | 222.44 (31.317) | 222.84 (25.395) | 245.94 (30.425) | 243.26 (21.967) | 244.19 (29.987) | 242.04 (22.956)
  Day 5: number analyzed (Participants) | 25 | 23 | 23 | 26 | 22 | 25 | 25 | 24 | 22
  Day 5 | 169.20 (28.586) | 154.83 (30.045) | 156.91 (22.240) | 219.42 (24.861) | 197.77 (25.487) | 211.56 (37.176) | 203.56 (28.777) | 199.58 (41.618) | 249.09 (24.156)
  Day 8: number analyzed (Participants) | 25 | 24 | 24 | 25 | 21 | 25 | 24 | 22 | 23
  Day 8 | 149.72 (24.979) | 137.71 (31.992) | 136.50 (21.364) | 222.68 (28.253) | 190.19 (20.856) | 202.44 (37.095) | 184.58 (30.935) | 186.73 (44.905) | 254.26 (22.481)
  Day 15 | 154.20 (26.011) | 137.83 (27.241) | 120.75 (25.589) | 221.69 (23.988) | 190.50 (20.964) | 198.64 (39.145) | 165.48 (30.456) | 165.71 (37.735) | 251.91 (24.830)
  Day 22: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 22 | 129.28 (22.856) | 119.00 (26.462) | 112.78 (19.247) | 218.12 (24.006) | 190.64 (23.768) | 176.28 (36.510) | 152.63 (29.854) | 153.67 (43.213) | 253.57 (15.716)
  Day 29: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 25 | 25 | 24 | 22
  Day 29 | 141.04 (27.355) | 133.54 (25.507) | 114.91 (24.487) | 217.12 (24.280) | 192.41 (31.173) | 176.36 (41.260) | 153.20 (25.762) | 150.42 (34.557) | 256.73 (22.391)
  Day 36: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 36 | 124.12 (22.380) | 113.88 (25.000) | 107.35 (19.590) | 217.08 (26.204) | 187.55 (30.803) | 163.48 (39.528) | 147.08 (25.568) | 144.63 (40.577) | 244.65 (24.356)
  Day 43 | 139.40 (23.944) | 128.83 (30.724) | 113.75 (23.167) | 214.62 (19.179) | 190.86 (28.734) | 171.96 (40.287) | 151.80 (23.638) | 147.25 (41.429) | 254.04 (19.793)
  Day 50: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Day 50 | 120.04 (20.687) | 112.63 (23.585) | 107.74 (22.471) | 215.42 (23.262) | 189.18 (24.209) | 161.00 (37.653) | 145.22 (24.814) | 144.17 (40.223) | 246.09 (17.776)
  Day 57: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 57 | 134.16 (25.826) | 116.96 (24.489) | 104.61 (20.045) | 208.04 (23.282) | 184.14 (31.148) | 158.96 (39.046) | 148.00 (30.107) | 135.83 (39.794) | 236.78 (16.105)
  Day 71: number analyzed (Participants) | 24 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 71 | 142.13 (29.489) | 121.04 (28.608) | 113.48 (25.056) | 218.38 (23.474) | 192.91 (31.288) | 174.64 (37.758) | 146.17 (29.736) | 142.42 (37.326) | 243.74 (24.849)
  Day 85: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Day 85 | 135.52 (25.161) | 119.58 (24.959) | 109.57 (27.611) | 208.88 (24.747) | 198.82 (36.000) | 165.44 (32.651) | 141.09 (31.318) | 134.17 (30.972) | 231.52 (22.701)
  Day 99: number analyzed (Participants) | 25 | 24 | 22 | 25 | 22 | 25 | 24 | 24 | 23
  Day 99 | 151.24 (31.139) | 128.58 (28.864) | 122.36 (36.702) | 216.28 (19.250) | 194.05 (33.230) | 178.36 (33.103) | 149.83 (33.780) | 139.13 (32.510) | 249.83 (19.277)
  Day 106: number analyzed (Participants) | 25 | 24 | 22 | 25 | 22 | 25 | 23 | 24 | 23
  Day 106 | 126.40 (29.017) | 114.75 (26.967) | 118.55 (29.987) | 212.36 (22.002) | 190.27 (28.352) | 167.84 (32.859) | 142.26 (32.265) | 139.92 (35.003) | 241.65 (18.982)
  Day 113: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 23 | 23
  Day 113 | 140.63 (26.650) | 124.58 (27.910) | 115.17 (30.293) | 201.64 (26.967) | 191.73 (34.189) | 169.72 (31.052) | 146.00 (33.889) | 134.17 (31.400) | 236.83 (16.808)
  Day 127: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 25 | 23 | 24 | 23
  Day 127 | 193.96 (26.253) | 176.88 (32.328) | 147.87 (37.486) | 219.32 (26.684) | 221.18 (32.444) | 223.16 (39.032) | 176.74 (46.917) | 166.63 (34.144) | 249.78 (25.598)
  Day 141: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 24 | 23
  Day 141 | 209.75 (32.446) | 202.71 (26.989) | 184.09 (38.141) | 216.48 (22.450) | 229.50 (38.480) | 247.36 (40.025) | 217.43 (43.351) | 192.96 (37.406) | 253.48 (21.494)
  Day 155: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 23 | 23 | 24 | 23
  Day 155 | 208.32 (28.912) | 203.83 (24.533) | 195.26 (31.865) | 221.28 (24.455) | 228.86 (37.640) | 250.00 (34.453) | 227.83 (31.438) | 208.25 (33.069) | 246.35 (15.171)
  Day 169: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 24 | 23 | 23 | 22
  Day 169 | 212.96 (29.508) | 212.79 (25.267) | 211.00 (31.348) | 221.00 (26.091) | 234.95 (43.216) | 254.17 (32.859) | 245.57 (34.103) | 227.65 (39.088) | 258.64 (20.537)

6. Secondary Outcome: Change From Baseline in Total Cholesterol (TC) at Day 85 and Day 113
Description: as for outcome 5
Time Frame: Baseline, Day 85, 113
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 26 | 22 | 25 | 25 | 24 | 23
mg/dL
  Change at Day 85: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Change at Day 85 | -78.64 (28.525) | -90.71 (31.705) | -101.43 (25.436) | -13.56 (22.346) | -24.02 (26.166) | -80.50 (31.851) | -102.80 (34.603) | -110.02 (24.119) | -10.52 (26.111)
  Change at Day 113: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 23 | 23
  Change at Day 113 | -73.44 (21.242) | -85.71 (30.263) | -95.83 (27.765) | -21.68 (23.686) | -31.11 (24.992) | -76.22 (36.301) | -97.89 (29.274) | -111.96 (24.871) | -5.22 (20.333)
Statistical Analysis 1: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-value (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -69.537, 95% CI 2-sided [-80.900 to -58.175], Standard Error of Mean 5.721
Statistical Analysis 2: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -86.446, 95% CI 2-sided [-98.074 to -74.818], Standard Error of Mean 5.855
Statistical Analysis 3: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -98.273, 95% CI 2-sided [-109.983 to -86.563], Standard Error of Mean 5.898
Statistical Analysis 4: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -71.435, 95% CI 2-sided [-85.757 to -57.112], Standard Error of Mean 7.209
Statistical Analysis 5: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -94.959, 95% CI 2-sided [-109.333 to -80.585], Standard Error of Mean 7.236
Statistical Analysis 6: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -98.519, 95% CI 2-sided [-112.727 to -84.311], Standard Error of Mean 7.150
Statistical Analysis 7: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -55.191, 95% CI 2-sided [-66.592 to -43.791], Standard Error of Mean 5.741
Statistical Analysis 8: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -72.211, 95% CI 2-sided [-83.825 to -60.597], Standard Error of Mean 5.848
Statistical Analysis 9: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -83.065, 95% CI 2-sided [-94.807 to -71.323], Standard Error of Mean 5.913
Statistical Analysis 10: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -73.879, 95% CI 2-sided [-87.147 to -60.612], Standard Error of Mean 6.678
Statistical Analysis 11: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -95.428, 95% CI 2-sided [-108.732 to -82.124], Standard Error of Mean 6.697
Statistical Analysis 12: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -104.859, 95% CI 2-sided [-118.079 to -91.639], Standard Error of Mean 6.654

7. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (TC) at Day 85 and Day 113
Description: Total cholesterol is the sum of all the cholesterol within the blood. Fasting was required at least 10 hours before blood sample collection. Baseline was defined as the mean of the last two non-missing measurements collected prior to the first dose of study treatment. Both measurements must be within 10 days prior to the first dose of study treatment; if only one measurement was available 10 days prior to the first dose of study treatment, then that measurement served as the baseline value. Percent change from baseline = ([observed value divided by baseline value] minus 1) multiplied by 100.
Time Frame: Baseline, Day 85, 113
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 26 | 22 | 25 | 25 | 24 | 23
percent change
  Change at Day 85: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Change at Day 85 | -36.26 (11.313) | -42.64 (13.310) | -48.22 (11.066) | -5.47 (9.038) | -10.85 (11.295) | -32.56 (12.011) | -41.98 (12.224) | -45.28 (9.539) | -3.82 (10.484)
  Change at Day 113: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 23 | 23
  Change at Day 113 | -34.28 (8.799) | -40.55 (13.471) | -45.58 (12.422) | -9.18 (9.204) | -14.02 (10.900) | -30.50 (13.212) | -40.27 (11.798) | -45.71 (9.786) | -1.62 (8.941)
Statistical Analysis 1: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -31.642, 95% CI 2-sided [-37.039 to -26.246], Standard Error of Mean 2.717
Statistical Analysis 2: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -39.880, 95% CI 2-sided [-45.403 to -34.358], Standard Error of Mean 2.781
Statistical Analysis 3: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -45.889, 95% CI 2-sided [-51.450 to -40.329], Standard Error of Mean 2.800
Statistical Analysis 4: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -30.137, 95% CI 2-sided [-36.110 to -24.164], Standard Error of Mean 3.006
Statistical Analysis 5: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -39.525, 95% CI 2-sided [-45.520 to -33.531], Standard Error of Mean 3.018
Statistical Analysis 6: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -41.372, 95% CI 2-sided [-47.299 to -35.445], Standard Error of Mean 2.983
Statistical Analysis 7: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -25.374, 95% CI 2-sided [-30.717 to -20.032], Standard Error of Mean 2.690
Statistical Analysis 8: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -33.490, 95% CI 2-sided [-38.934 to -28.047], Standard Error of Mean 2.741
Statistical Analysis 9: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -38.760, 95% CI 2-sided [-44.262 to -33.258], Standard Error of Mean 2.770
Statistical Analysis 10: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -30.847, 95% CI 2-sided [-36.568 to -25.127], Standard Error of Mean 2.879
Statistical Analysis 11: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -40.019, 95% CI 2-sided [-45.754 to -34.285], Standard Error of Mean 2.887
Statistical Analysis 12: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 12]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -43.947, 95% CI 2-sided [-49.647 to -38.247], Standard Error of Mean 2.869

8. Secondary Outcome: Apolipoprotein B (ApoB)
Description: ApoB is a major protein that makes up LDL cholesterol and is involved in transporting cholesterol and triglycerides to cells and tissues in the body. Fasting was required at least 10 hours before blood sample collection. Baseline was defined as the mean of the last two non-missing measurements collected prior to the first dose of study treatment. Both measurements must be within 10 days prior to the first dose of study treatment; if only one measurement was available 10 days prior to the first dose of study treatment, then that measurement served as the baseline value.
Time Frame: Baseline, Day 5, 8, 15, 22, 29, 36, 43, 50, 57, 71, 85, 99, 106, 113, 127, 141, 155, 169
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 26 | 22 | 25 | 25 | 24 | 23
mg/dL
  Baseline | 92.76 (14.383) | 92.54 (12.362) | 90.40 (12.732) | 95.65 (13.229) | 96.70 (13.382) | 106.54 (15.800) | 104.02 (14.652) | 101.88 (11.494) | 103.13 (13.608)
  Day 5: number analyzed (Participants) | 25 | 23 | 23 | 26 | 22 | 25 | 25 | 24 | 22
  Day 5 | 67.72 (15.175) | 59.83 (14.269) | 60.26 (8.853) | 94.62 (12.847) | 84.68 (13.570) | 88.40 (18.777) | 82.88 (13.179) | 78.00 (14.025) | 104.86 (11.902)
  Day 8: number analyzed (Participants) | 25 | 24 | 24 | 25 | 21 | 25 | 24 | 22 | 23
  Day 8 | 56.12 (12.245) | 49.04 (15.982) | 47.42 (9.050) | 95.72 (16.395) | 80.38 (13.113) | 82.52 (19.402) | 71.71 (13.614) | 70.27 (16.237) | 107.61 (11.357)
  Day 15 | 60.20 (15.658) | 49.38 (15.528) | 36.50 (8.703) | 96.65 (13.069) | 79.36 (9.639) | 82.24 (21.127) | 62.28 (16.403) | 58.08 (12.265) | 107.39 (12.052)
  Day 22: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 22 | 44.28 (13.227) | 36.83 (12.923) | 31.09 (5.938) | 96.35 (10.954) | 79.77 (12.976) | 68.76 (20.949) | 53.46 (14.700) | 50.54 (15.300) | 108.35 (10.530)
  Day 29: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 25 | 25 | 24 | 22
  Day 29 | 52.08 (16.595) | 46.42 (16.264) | 32.83 (8.611) | 96.00 (11.800) | 80.73 (12.691) | 69.32 (20.613) | 54.20 (12.285) | 50.25 (11.752) | 107.23 (12.134)
  Day 36: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 36 | 41.04 (11.998) | 35.50 (13.603) | 29.43 (6.036) | 96.27 (14.717) | 80.18 (13.828) | 62.40 (19.885) | 49.25 (8.115) | 46.92 (14.191) | 103.74 (13.363)
  Day 43 | 51.36 (14.494) | 42.50 (17.942) | 31.96 (7.538) | 94.31 (9.216) | 82.68 (12.797) | 67.24 (19.959) | 53.60 (14.283) | 48.50 (14.301) | 110.39 (11.645)
  Day 50: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Day 50 | 38.48 (10.759) | 34.08 (12.728) | 30.52 (6.660) | 95.69 (12.802) | 82.86 (12.822) | 62.28 (19.932) | 49.43 (11.469) | 47.58 (14.443) | 107.22 (11.062)
  Day 57: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 57 | 49.44 (14.077) | 38.29 (16.236) | 29.48 (6.052) | 93.81 (12.316) | 79.68 (15.490) | 62.00 (19.660) | 53.25 (17.745) | 45.79 (12.322) | 104.13 (9.057)
  Day 71: number analyzed (Participants) | 24 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 71 | 52.83 (16.903) | 38.71 (16.648) | 32.00 (7.634) | 97.23 (11.884) | 85.18 (14.378) | 69.96 (19.673) | 50.63 (11.568) | 47.79 (12.112) | 107.78 (16.082)
  Day 85: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Day 85 | 51.32 (15.258) | 39.21 (15.291) | 33.65 (14.717) | 93.46 (12.666) | 86.77 (16.934) | 68.68 (17.409) | 49.35 (15.183) | 45.13 (10.678) | 102.09 (12.387)
  Day 99: number analyzed (Participants) | 25 | 24 | 22 | 25 | 22 | 25 | 24 | 24 | 23
  Day 99 | 57.36 (17.291) | 44.29 (17.853) | 37.55 (18.913) | 95.08 (12.165) | 84.05 (16.247) | 72.56 (18.063) | 53.63 (17.272) | 45.88 (11.211) | 110.91 (11.049)
  Day 106: number analyzed (Participants) | 25 | 24 | 22 | 25 | 22 | 25 | 23 | 24 | 23
  Day 106 | 42.12 (13.233) | 34.71 (15.029) | 35.55 (15.987) | 94.36 (12.192) | 83.32 (14.965) | 66.72 (17.111) | 48.87 (13.168) | 47.00 (12.332) | 107.48 (10.117)
  Day 113: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 23 | 23
  Day 113 | 53.50 (13.593) | 42.83 (16.612) | 36.48 (15.111) | 88.40 (13.438) | 82.77 (15.593) | 69.08 (17.007) | 52.52 (15.774) | 45.87 (11.530) | 105.61 (9.940)
  Day 127: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 25 | 23 | 24 | 23
  Day 127 | 82.00 (13.871) | 73.04 (21.566) | 54.61 (24.203) | 95.16 (12.216) | 98.50 (16.280) | 97.20 (20.827) | 69.91 (28.257) | 62.75 (19.525) | 111.35 (14.288)
  Day 141: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 24 | 23
  Day 141 | 89.50 (14.611) | 87.71 (18.112) | 74.87 (25.118) | 95.08 (12.024) | 100.45 (19.043) | 108.96 (21.279) | 92.70 (27.420) | 77.67 (25.466) | 110.09 (12.109)
  Day 155: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 23 | 23 | 24 | 23
  Day 155 | 90.16 (14.291) | 89.00 (15.836) | 81.87 (16.652) | 96.00 (11.832) | 101.23 (18.619) | 111.39 (17.758) | 98.26 (19.262) | 86.04 (23.451) | 108.43 (10.422)
  Day 169: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 24 | 23 | 23 | 22
  Day 169 | 93.36 (16.176) | 93.63 (14.455) | 91.57 (15.147) | 96.88 (13.532) | 103.09 (20.718) | 112.46 (16.005) | 105.91 (17.661) | 95.74 (21.764) | 111.41 (9.879)

9. Secondary Outcome: Change From Baseline in Apolipoprotein B (ApoB) at Day 85 and Day 113
Description: ApoB is a major protein that makes up LDL cholesterol and is involved in transporting cholesterol and triglycerides to cells and tissues in the body. Fasting was required at least 10 hours before blood sample collection. Baseline was defined as the mean of the last two non-missing measurements collected prior to the first dose of study treatment. Both measurements must be within 10 days prior to the first dose of study treatment; if only one measurement was available 10 days prior to the first dose of study treatment, then that measurement served as the baseline value. Change from baseline = observed value minus baseline value.
Time Frame: Baseline, Day 85, 113
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 26 | 22 | 25 | 25 | 24 | 23
mg/dL
  Change at Day 85: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Change at Day 85 | -41.44 (16.385) | -53.33 (19.097) | -56.43 (17.650) | -2.19 (10.703) | -9.93 (14.350) | -37.86 (18.125) | -54.33 (21.080) | -56.75 (14.506) | -1.04 (13.020)
  Change at Day 113: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 23 | 23
  Change at Day 113 | -39.56 (12.011) | -49.71 (18.699) | -53.61 (16.526) | -7.70 (12.436) | -13.93 (12.650) | -37.46 (18.504) | -51.15 (16.855) | -56.83 (15.501) | 2.48 (11.107)
Statistical Analysis 1: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -41.118, 95% CI 2-sided [-47.760 to -34.476], Standard Error of Mean 3.344
Statistical Analysis 2: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -54.787, 95% CI 2-sided [-61.543 to -48.032], Standard Error of Mean 3.402
Statistical Analysis 3: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -60.549, 95% CI 2-sided [-67.403 to -53.694], Standard Error of Mean 3.453
Statistical Analysis 4: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -36.589, 95% CI 2-sided [-43.999 to -29.178], Standard Error of Mean 3.730
Statistical Analysis 5: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -54.683, 95% CI 2-sided [-62.102 to -47.265], Standard Error of Mean 3.734
Statistical Analysis 6: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -56.517, 95% CI 2-sided [-63.845 to -49.189], Standard Error of Mean 3.688
Statistical Analysis 7: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -33.262, 95% CI 2-sided [-39.608 to -26.915], Standard Error of Mean 3.196
Statistical Analysis 8: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -45.956, 95% CI 2-sided [-52.388 to -39.523], Standard Error of Mean 3.239
Statistical Analysis 9: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -51.500, 95% CI 2-sided [-58.063 to -44.937], Standard Error of Mean 3.305
Statistical Analysis 10: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -40.474, 95% CI 2-sided [-47.523 to -33.426], Standard Error of Mean 3.547
Statistical Analysis 11: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -54.634, 95% CI 2-sided [-61.685 to -47.583], Standard Error of Mean 3.549
Statistical Analysis 12: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 12]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -59.608, 95% CI 2-sided [-66.602 to -52.614], Standard Error of Mean 3.520

10. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B (ApoB) at Day 85 and Day 113
Description: ApoB is a major protein that makes up LDL cholesterol and is involved in transporting cholesterol and triglycerides to cells and tissues in the body. Fasting was required at least 10 hours before blood sample collection. Baseline was defined as the mean of the last two non-missing measurements collected prior to the first dose of study treatment. Both measurements must be within 10 days prior to the first dose of study treatment; if only one measurement was available 10 days prior to the first dose of study treatment, then that measurement served as the baseline value. Percent change from baseline = ([observed value divided by baseline value] minus 1) multiplied by 100.
Time Frame: Baseline, Day 85, 113
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 26 | 22 | 25 | 25 | 24 | 23
percent change
  Change at Day 85: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Change at Day 85 | -44.30 (15.675) | -57.02 (17.985) | -62.31 (15.684) | -1.77 (10.567) | -9.97 (14.426) | -35.16 (15.906) | -51.62 (16.289) | -55.31 (11.060) | -0.13 (12.144)
  Change at Day 113: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 23 | 23
  Change at Day 113 | -42.64 (11.864) | -53.45 (18.449) | -59.48 (15.320) | -7.54 (11.662) | -14.17 (12.713) | -34.66 (16.214) | -49.10 (14.474) | -54.88 (12.109) | 3.43 (12.038)
Statistical Analysis 1: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -43.265, 95% CI 2-sided [-50.347 to -36.183], Standard Error of Mean 3.566
Statistical Analysis 2: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -57.962, 95% CI 2-sided [-65.167 to -50.758], Standard Error of Mean 3.628
Statistical Analysis 3: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -64.729, 95% CI 2-sided [-72.039 to -57.419], Standard Error of Mean 3.682
Statistical Analysis 4: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -36.428, 95% CI 2-sided [-43.451 to -29.405], Standard Error of Mean 3.535
Statistical Analysis 5: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -53.296, 95% CI 2-sided [-60.325 to -46.267], Standard Error of Mean 3.538
Statistical Analysis 6: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -55.489, 95% CI 2-sided [-62.436 to -48.542], Standard Error of Mean 3.496
Statistical Analysis 7: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -35.288, 95% CI 2-sided [-42.059 to -28.516], Standard Error of Mean 3.410
Statistical Analysis 8: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -48.845, 95% CI 2-sided [-55.709 to -41.982], Standard Error of Mean 3.456
Statistical Analysis 9: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -55.114, 95% CI 2-sided [-62.116 to -48.112], Standard Error of Mean 3.526
Statistical Analysis 10: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -40.045, 95% CI 2-sided [-47.118 to -32.971], Standard Error of Mean 3.560
Statistical Analysis 11: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -53.810, 95% CI 2-sided [-60.883 to -46.737], Standard Error of Mean 3.560
Statistical Analysis 12: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 12]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -58.620, 95% CI 2-sided [-65.640 to -51.600], Standard Error of Mean 3.533

11. Secondary Outcome: Apolipoprotein A-I (ApoA-I)
Description: ApoA1 is a major protein that is a component of HDL cholesterol and helps in clearing cholesterol from the blood by removing cholesterol from organs and tissues to be destroyed by the liver. Fasting was required at least 10 hours before blood sample collection. Baseline was defined as the mean of the last two non-missing measurements collected prior to the first dose of study treatment. Both measurements must be within 10 days prior to the first dose of study treatment; if only one measurement was available 10 days prior to the first dose of study treatment, then that measurement served as the baseline value.
Time Frame: Baseline, Day 5, 8, 15, 22, 29, 36, 43, 50, 57, 71, 85, 99, 106, 113, 127, 141, 155, 169
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 26 | 22 | 25 | 25 | 24 | 23
mg/dL
  Baseline | 137.02 (13.235) | 142.60 (16.507) | 140.31 (18.813) | 145.65 (21.908) | 145.34 (16.171) | 138.90 (21.808) | 145.38 (19.260) | 146.75 (25.587) | 150.13 (16.834)
  Day 5: number analyzed (Participants) | 25 | 23 | 23 | 26 | 22 | 25 | 25 | 24 | 22
  Day 5 | 140.72 (14.644) | 146.65 (16.773) | 144.48 (19.943) | 146.08 (21.505) | 144.68 (16.193) | 142.12 (22.260) | 145.12 (18.485) | 149.79 (24.285) | 150.09 (17.989)
  Day 8: number analyzed (Participants) | 25 | 24 | 24 | 25 | 21 | 25 | 24 | 22 | 23
  Day 8 | 140.44 (14.972) | 147.46 (16.707) | 146.88 (19.200) | 147.00 (21.527) | 145.57 (16.351) | 146.76 (25.406) | 145.79 (19.260) | 152.45 (28.118) | 150.48 (16.782)
  Day 15 | 141.56 (13.811) | 153.00 (16.325) | 150.46 (20.479) | 147.04 (22.704) | 148.50 (18.918) | 145.76 (23.197) | 150.08 (20.762) | 157.04 (25.154) | 151.00 (19.214)
  Day 22: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 22 | 143.20 (15.554) | 152.88 (18.473) | 151.78 (20.576) | 145.31 (21.481) | 146.41 (17.012) | 145.96 (22.354) | 150.08 (19.019) | 155.17 (23.265) | 151.65 (17.185)
  Day 29: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 25 | 25 | 24 | 22
  Day 29 | 144.32 (15.118) | 155.79 (19.598) | 151.78 (22.913) | 144.28 (20.633) | 146.23 (17.221) | 146.36 (22.503) | 150.04 (21.763) | 155.96 (23.143) | 154.32 (15.304)
  Day 36: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 36 | 143.48 (15.273) | 149.88 (17.957) | 150.13 (21.102) | 143.46 (20.609) | 145.91 (18.652) | 145.08 (22.953) | 153.33 (19.417) | 155.08 (24.063) | 149.30 (18.639)
  Day 43 | 144.52 (12.842) | 153.88 (18.262) | 150.33 (22.584) | 142.42 (21.495) | 144.64 (16.105) | 146.00 (21.050) | 152.32 (21.059) | 155.75 (32.193) | 149.04 (16.932)
  Day 50: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Day 50 | 145.80 (15.042) | 151.25 (19.157) | 149.13 (19.008) | 143.46 (20.397) | 141.95 (15.807) | 142.84 (21.885) | 152.52 (19.739) | 153.92 (25.100) | 145.70 (14.348)
  Day 57: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 57 | 138.40 (14.919) | 149.46 (19.509) | 145.83 (18.930) | 137.62 (18.206) | 142.18 (15.445) | 136.32 (20.010) | 145.96 (22.029) | 144.96 (25.049) | 138.87 (16.491)
  Day 71: number analyzed (Participants) | 24 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 71 | 145.50 (16.192) | 152.92 (21.086) | 150.43 (21.002) | 142.62 (19.150) | 144.18 (15.383) | 143.88 (21.896) | 151.88 (17.523) | 154.25 (23.130) | 146.17 (14.981)
  Day 85: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Day 85 | 138.04 (14.968) | 148.17 (16.818) | 144.04 (15.933) | 136.00 (20.229) | 144.23 (14.498) | 132.88 (19.303) | 145.13 (17.168) | 146.58 (23.006) | 136.30 (16.753)
  Day 99: number analyzed (Participants) | 25 | 24 | 22 | 25 | 22 | 25 | 24 | 24 | 23
  Day 99 | 147.40 (18.771) | 154.54 (17.840) | 150.86 (21.108) | 147.48 (20.799) | 145.91 (16.798) | 143.88 (19.577) | 151.29 (21.612) | 149.83 (20.750) | 144.65 (19.812)
  Day 106: number analyzed (Participants) | 25 | 24 | 22 | 25 | 22 | 25 | 23 | 24 | 23
  Day 106 | 145.92 (18.773) | 154.96 (19.282) | 150.23 (18.341) | 143.12 (17.822) | 144.64 (15.413) | 142.56 (21.143) | 149.26 (19.909) | 150.46 (21.444) | 141.17 (15.497)
  Day 113: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 23 | 23
  Day 113 | 139.21 (15.731) | 149.17 (18.719) | 144.13 (18.587) | 137.72 (21.454) | 145.00 (14.690) | 138.40 (19.581) | 149.09 (18.033) | 143.96 (21.353) | 140.04 (16.767)
  Day 127: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 25 | 23 | 24 | 23
  Day 127 | 144.08 (18.630) | 148.75 (17.738) | 150.04 (23.145) | 145.60 (22.763) | 144.27 (14.701) | 141.68 (20.412) | 148.48 (18.012) | 149.17 (23.566) | 144.48 (15.237)
  Day 141: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 24 | 23
  Day 141 | 145.46 (19.006) | 151.21 (18.990) | 154.17 (22.321) | 148.52 (23.261) | 144.45 (16.721) | 141.36 (20.968) | 148.74 (17.324) | 151.29 (22.831) | 149.13 (19.328)
  Day 155: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 23 | 23 | 24 | 23
  Day 155 | 143.52 (17.564) | 148.83 (20.267) | 149.52 (21.848) | 147.60 (23.076) | 147.09 (16.446) | 140.96 (23.437) | 148.09 (21.037) | 149.13 (23.899) | 148.83 (18.077)
  Day 169: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 24 | 23 | 23 | 22
  Day 169 | 142.96 (20.387) | 151.54 (19.010) | 150.96 (19.025) | 154.88 (23.938) | 153.64 (21.367) | 144.13 (24.746) | 151.70 (21.699) | 151.13 (29.425) | 154.36 (19.742)

12. Secondary Outcome: Change From Baseline in Apolipoprotein A-I (ApoA-I) at Day 85 and Day 113
Description: ApoA1 is a major protein that is a component of HDL cholesterol and helps in clearing cholesterol from the blood by removing cholesterol from organs and tissues to be destroyed by the liver. Fasting was required at least 10 hours before blood sample collection. Baseline was defined as the mean of the last two non-missing measurements collected prior to the first dose of study treatment. Both measurements must be within 10 days prior to the first dose of study treatment; if only one measurement was available 10 days prior to the first dose of study treatment, then that measurement served as the baseline value. Change from baseline = observed value minus baseline value.
Time Frame: Baseline, Day 85, 113
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 26 | 22 | 25 | 25 | 24 | 23
mg/dL
  Change at Day 85: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Change at Day 85 | 1.02 (9.479) | 5.56 (10.575) | 3.63 (11.155) | -9.65 (9.495) | -1.11 (11.118) | -6.02 (11.069) | -2.09 (12.040) | -0.17 (11.897) | -13.83 (10.602)
  Change at Day 113: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 23 | 23
  Change at Day 113 | 2.52 (9.226) | 6.56 (12.310) | 3.72 (11.977) | -7.86 (13.052) | -0.34 (10.783) | -0.50 (9.512) | 1.87 (9.328) | -3.54 (8.982) | -10.09 (11.236)
Statistical Analysis 1: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 8.896, 95% CI 2-sided [3.646 to 14.145], Standard Error of Mean 2.643
Statistical Analysis 2: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 15.429, 95% CI 2-sided [10.141 to 20.717], Standard Error of Mean 2.662
Statistical Analysis 3: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 12.321, 95% CI 2-sided [6.959 to 17.683], Standard Error of Mean 2.700
Statistical Analysis 4: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.014, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 6.804, 95% CI 2-sided [0.761 to 12.847], Standard Error of Mean 3.041
Statistical Analysis 5: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 10.565, 95% CI 2-sided [4.556 to 16.573], Standard Error of Mean 3.023
Statistical Analysis 6: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 12.895, 95% CI 2-sided [6.993 to 18.796], Standard Error of Mean 2.969
Statistical Analysis 7: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 8.644, 95% CI 2-sided [2.157 to 15.130], Standard Error of Mean 3.266
Statistical Analysis 8: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 14.708, 95% CI 2-sided [8.208 to 21.208], Standard Error of Mean 3.272
Statistical Analysis 9: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 11.168, 95% CI 2-sided [4.580 to 17.757], Standard Error of Mean 3.317
Statistical Analysis 10: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 8.132, 95% CI 2-sided [2.947 to 13.316], Standard Error of Mean 2.609
Statistical Analysis 11: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 10.230, 95% CI 2-sided [5.079 to 15.381], Standard Error of Mean 2.592
Statistical Analysis 12: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 12]; Test type: Superiority or Other; p = 0.014, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 5.767, 95% CI 2-sided [0.670 to 10.864], Standard Error of Mean 2.565

13. Secondary Outcome: Percent Change From Baseline in Apolipoprotein A-I (ApoA-I) at Day 85 and Day 113
Description: ApoA1 is a major protein that is a component of HDL cholesterol and helps in clearing cholesterol from the blood by removing cholesterol from organs and tissues to be destroyed by the liver. Fasting was required at least 10 hours before blood sample collection. Baseline was defined as the mean of the last two non-missing measurements collected prior to the first dose of study treatment. Both measurements must be within 10 days prior to the first dose of study treatment; if only one measurement was available 10 days prior to the first dose of study treatment, then that measurement served as the baseline value. Percent change from baseline = ([observed value divided by baseline value] minus 1) multiplied by 100.
Time Frame: Baseline, Day 85, 113
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 26 | 22 | 25 | 25 | 24 | 23
percent change
  Change at Day 85: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Change at Day 85 | 0.87 (7.002) | 4.20 (7.438) | 3.26 (8.418) | -6.44 (6.252) | -0.34 (7.749) | -3.82 (8.033) | -1.00 (8.245) | 0.44 (8.673) | -9.10 (6.738)
  Change at Day 113: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 23 | 23
  Change at Day 113 | 1.93 (6.789) | 4.82 (8.766) | 3.13 (8.663) | -5.16 (8.106) | 0.15 (7.819) | 0.13 (7.013) | 1.53 (6.572) | -1.84 (5.923) | -6.55 (6.903)
Statistical Analysis 1: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 6.079, 95% CI 2-sided [2.296 to 9.863], Standard Error of Mean 1.905
Statistical Analysis 2: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 10.786, 95% CI 2-sided [6.976 to 14.597], Standard Error of Mean 1.918
Statistical Analysis 3: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 9.069, 95% CI 2-sided [5.206 to 12.932], Standard Error of Mean 1.945
Statistical Analysis 4: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.014, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 4.859, 95% CI 2-sided [0.541 to 9.178], Standard Error of Mean 2.173
Statistical Analysis 5: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 7.331, 95% CI 2-sided [3.037 to 11.624], Standard Error of Mean 2.161
Statistical Analysis 6: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 9.075, 95% CI 2-sided [4.856 to 13.293], Standard Error of Mean 2.122
Statistical Analysis 7: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 5.936, 95% CI 2-sided [1.435 to 10.437], Standard Error of Mean 2.266
Statistical Analysis 8: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 10.213, 95% CI 2-sided [5.702 to 14.724], Standard Error of Mean 2.271
Statistical Analysis 9: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 8.056, 95% CI 2-sided [3.484 to 12.629], Standard Error of Mean 2.302
Statistical Analysis 10: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 5.846, 95% CI 2-sided [2.312 to 9.380], Standard Error of Mean 1.778
Statistical Analysis 11: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 6.910, 95% CI 2-sided [3.400 to 10.421], Standard Error of Mean 1.766
Statistical Analysis 12: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 12]; Test type: Superiority or Other; p = 0.010, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 4.168, 95% CI 2-sided [0.693 to 7.642], Standard Error of Mean 1.748

14. Secondary Outcome: Apolipoprotein A-II (ApoA-II)
Description: ApoA-II is the second most abundant component of the HDL cholesterol. Fasting was required at least 10 hours before blood sample collection. Baseline was defined as the mean of the last two non-missing measurements collected prior to the first dose of study treatment. Both measurements must be within 10 days prior to the first dose of study treatment; if only one measurement was available 10 days prior to the first dose of study treatment, then that measurement served as the baseline value.
Time Frame: Baseline, Day 5, 8, 15, 22, 29, 36, 43, 50, 57, 71, 85, 99, 106, 113, 127, 141, 155, 169
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 26 | 22 | 25 | 25 | 24 | 23
mg/dL
  Baseline | 30.700 (3.6817) | 30.223 (2.8992) | 30.471 (2.8918) | 31.515 (3.8373) | 32.189 (3.2855) | 29.940 (3.3630) | 31.232 (3.9681) | 30.294 (3.0541) | 31.354 (3.9552)
  Day 5: number analyzed (Participants) | 25 | 23 | 23 | 26 | 22 | 25 | 25 | 24 | 22
  Day 5 | 30.884 (3.6551) | 30.161 (2.9004) | 30.443 (3.4057) | 31.608 (3.6099) | 32.709 (3.4130) | 30.088 (3.4784) | 30.972 (4.2462) | 30.558 (3.0567) | 31.473 (4.1750)
  Day 8: number analyzed (Participants) | 25 | 24 | 24 | 25 | 21 | 25 | 24 | 22 | 23
  Day 8 | 30.224 (2.8736) | 30.675 (3.1077) | 30.738 (2.9137) | 32.036 (3.2261) | 32.495 (3.0372) | 30.760 (3.3363) | 30.608 (3.8492) | 30.664 (3.2942) | 31.635 (3.6272)
  Day 15 | 30.528 (3.7034) | 31.129 (2.9304) | 31.304 (3.0309) | 32.062 (3.2968) | 33.136 (3.6822) | 30.568 (3.3308) | 31.516 (3.9116) | 31.275 (3.4925) | 31.530 (4.6451)
  Day 22: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 22 | 31.232 (3.1787) | 30.667 (3.4561) | 31.183 (3.8763) | 31.846 (3.0899) | 32.273 (3.2310) | 30.620 (3.3448) | 31.125 (4.0921) | 30.896 (3.0900) | 32.200 (3.6940)
  Day 29: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 25 | 25 | 24 | 22
  Day 29 | 31.608 (3.2712) | 32.279 (4.1331) | 31.035 (3.7585) | 32.096 (3.6363) | 32.395 (3.1748) | 30.740 (3.0899) | 31.100 (3.6272) | 31.071 (2.8639) | 31.882 (3.6960)
  Day 36: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 36 | 31.208 (3.5747) | 30.838 (3.3920) | 30.622 (3.3870) | 31.150 (3.3011) | 32.091 (4.0243) | 29.768 (3.2825) | 31.404 (4.0581) | 30.975 (3.3526) | 31.478 (3.7066)
  Day 43 | 31.600 (3.8155) | 31.908 (4.2809) | 31.004 (3.6090) | 31.685 (3.6743) | 32.636 (3.1568) | 30.720 (3.6371) | 32.408 (4.0300) | 31.138 (3.4691) | 31.922 (3.8381)
  Day 50: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Day 50 | 31.772 (3.9676) | 31.117 (3.5511) | 30.991 (2.9264) | 31.900 (3.5621) | 32.282 (3.5327) | 29.760 (3.8077) | 32.704 (3.8668) | 31.083 (3.8423) | 30.830 (3.7644)
  Day 57: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 57 | 30.708 (5.1285) | 30.271 (4.0390) | 29.987 (3.2086) | 30.773 (3.4292) | 32.405 (3.0798) | 28.548 (3.8710) | 31.454 (4.3687) | 30.033 (3.9031) | 29.861 (3.3007)
  Day 71: number analyzed (Participants) | 24 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 71 | 32.600 (4.3091) | 31.554 (4.3823) | 31.148 (2.8016) | 32.092 (3.5748) | 33.127 (3.3208) | 30.260 (3.9125) | 32.658 (3.9677) | 31.804 (3.5119) | 31.317 (4.0283)
  Day 85: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Day 85 | 30.484 (4.5441) | 30.296 (4.2019) | 29.974 (3.3766) | 30.577 (4.1019) | 33.095 (3.4642) | 29.036 (3.6811) | 31.957 (4.8917) | 30.533 (4.0376) | 29.657 (3.6082)
  Day 99: number analyzed (Participants) | 25 | 24 | 22 | 25 | 22 | 25 | 24 | 24 | 23
  Day 99 | 32.868 (4.2145) | 32.054 (4.3729) | 31.436 (3.7821) | 32.500 (4.3987) | 33.155 (3.9087) | 31.352 (3.8161) | 32.925 (5.9562) | 31.229 (2.9670) | 31.570 (4.3204)
  Day 106: number analyzed (Participants) | 25 | 24 | 22 | 25 | 22 | 25 | 23 | 24 | 23
  Day 106 | 31.908 (4.1181) | 31.850 (3.8284) | 31.073 (3.3504) | 31.724 (3.5444) | 32.432 (3.6429) | 30.520 (3.9332) | 32.552 (4.3131) | 31.438 (3.7623) | 30.865 (3.7092)
  Day 113: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 23 | 23
  Day 113 | 30.442 (4.1097) | 30.313 (4.1545) | 29.787 (3.3975) | 30.388 (3.3572) | 32.559 (3.0055) | 29.300 (3.3821) | 32.361 (4.1480) | 30.239 (3.2747) | 30.126 (3.5101)
  Day 127: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 25 | 23 | 24 | 23
  Day 127 | 32.068 (3.9869) | 31.358 (3.9263) | 31.370 (3.4158) | 31.824 (3.4922) | 32.905 (3.2614) | 30.904 (3.1115) | 32.374 (3.7973) | 31.242 (3.5215) | 31.839 (3.7256)
  Day 141: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 24 | 23
  Day 141 | 32.704 (4.5005) | 32.325 (4.2787) | 32.835 (3.3582) | 32.044 (4.2146) | 32.818 (3.4188) | 31.412 (3.6261) | 33.287 (3.0694) | 32.029 (3.4970) | 32.178 (3.1213)
  Day 155: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 23 | 23 | 24 | 23
  Day 155 | 32.164 (3.9476) | 31.629 (4.4463) | 31.878 (3.3637) | 31.956 (4.1374) | 32.877 (3.7858) | 31.061 (3.8024) | 32.891 (4.0870) | 31.867 (3.6487) | 31.439 (3.4050)
  Day 169: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 24 | 23 | 23 | 22
  Day 169 | 31.848 (4.1778) | 32.033 (3.8588) | 32.352 (3.8903) | 33.120 (4.2339) | 33.623 (4.2722) | 31.433 (3.8678) | 33.578 (4.4671) | 32.070 (3.9987) | 32.345 (3.6908)

15. Secondary Outcome: Change From Baseline in Apolipoprotein A-II (ApoA-II) at Day 85 and Day 113
Description: ApoA-II is the second most abundant component of the HDL cholesterol. Fasting was required at least 10 hours before blood sample collection. Baseline was defined as the mean of the last two non-missing measurements collected prior to the first dose of study treatment. Both measurements must be within 10 days prior to the first dose of study treatment; if only one measurement was available 10 days prior to the first dose of study treatment, then that measurement served as the baseline value. Change from baseline = observed value minus baseline value.
Time Frame: Baseline, Day 85, 113
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 26 | 22 | 25 | 25 | 24 | 23
mg/dL
  Change at Day 85: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Change at Day 85 | -0.216 (2.2274) | 0.073 (2.6605) | -0.450 (2.3906) | -0.938 (1.8339) | 0.907 (2.6785) | -0.904 (2.3894) | 0.354 (3.3769) | 0.240 (3.1812) | -1.698 (2.9589)
  Change at Day 113: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 23 | 23
  Change at Day 113 | -0.073 (2.0937) | 0.090 (2.3882) | -0.637 (2.2412) | -1.104 (4.0438) | 0.370 (2.2388) | -0.640 (2.0394) | 0.759 (2.2739) | 0.002 (2.8256) | -1.228 (3.4404)
Statistical Analysis 1: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.127, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 0.7208, 95% CI 2-sided [-0.5283 to 1.9700], Standard Error of Mean 0.6289
Statistical Analysis 2: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.053, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 1.0574, 95% CI 2-sided [-0.2259 to 2.3406], Standard Error of Mean 0.6461
Statistical Analysis 3: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.354, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 0.2445, 95% CI 2-sided [-1.0486 to 1.5375], Standard Error of Mean 0.6511
Statistical Analysis 4: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.176, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 0.8055, 95% CI 2-sided [-0.9066 to 2.5177], Standard Error of Mean 0.8615
Statistical Analysis 5: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.011, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 2.0071, 95% CI 2-sided [0.2899 to 3.7242], Standard Error of Mean 0.8641
Statistical Analysis 6: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.024, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 1.7116, 95% CI 2-sided [0.0184 to 3.4049], Standard Error of Mean 0.8520
Statistical Analysis 7: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.138, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 0.8585, 95% CI 2-sided [-0.6992 to 2.4163], Standard Error of Mean 0.7844
Statistical Analysis 8: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.137, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 0.8807, 95% CI 2-sided [-0.7064 to 2.4678], Standard Error of Mean 0.7990
Statistical Analysis 9: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.373, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 0.2624, 95% CI 2-sided [-1.3370 to 1.8618], Standard Error of Mean 0.8053
Statistical Analysis 10: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.333, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 0.3239, 95% CI 2-sided [-1.1611 to 1.8089], Standard Error of Mean 0.7472
Statistical Analysis 11: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.006, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 1.9322, 95% CI 2-sided [0.4441 to 3.4203], Standard Error of Mean 0.7488
Statistical Analysis 12: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 12]; Test type: Superiority or Other; p = 0.133, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 0.8340, 95% CI 2-sided [-0.6451 to 2.3130], Standard Error of Mean 0.7442

16. Secondary Outcome: Percent Change From Baseline in Apolipoprotein A-II (ApoA-II) at Day 85 and Day 113
Description: ApoA-II is the second most abundant component of the HDL cholesterol. Fasting was required at least 10 hours before blood sample collection. Baseline was defined as the mean of the last two non-missing measurements collected prior to the first dose of study treatment. Both measurements must be within 10 days prior to the first dose of study treatment; if only one measurement was available 10 days prior to the first dose of study treatment, then that measurement served as the baseline value. Percent change from baseline = ([observed value divided by baseline value] minus 1) multiplied by 100.
Time Frame: Baseline, Day 85, 113
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 26 | 22 | 25 | 25 | 24 | 23
percent change
  Change at Day 85: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Change at Day 85 | -0.85 (7.387) | 0.17 (8.699) | -1.34 (7.672) | -2.93 (5.741) | 3.13 (8.288) | -2.87 (7.788) | 1.34 (10.779) | 0.98 (10.565) | -4.97 (9.262)
  Change at Day 113: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 23 | 23
  Change at Day 113 | -0.21 (6.972) | 0.13 (7.974) | -1.99 (7.403) | -2.77 (11.234) | 1.48 (6.776) | -1.94 (6.337) | 2.64 (7.315) | 0.39 (9.526) | -3.29 (10.137)
Statistical Analysis 1: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.155, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 2.0813, 95% CI 2-sided [-1.9730 to 6.1356], Standard Error of Mean 2.0411
Statistical Analysis 2: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.062, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 3.2608, 95% CI 2-sided [-0.9035 to 7.4250], Standard Error of Mean 2.0965
Statistical Analysis 3: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.349, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 0.8224, 95% CI 2-sided [-3.3733 to 5.0182], Standard Error of Mean 2.1126
Statistical Analysis 4: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.202, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 2.3254, 95% CI 2-sided [-3.1801 to 7.8310], Standard Error of Mean 2.7702
Statistical Analysis 5: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.015, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 6.1048, 95% CI 2-sided [0.5833 to 11.6263], Standard Error of Mean 2.7784
Statistical Analysis 6: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.030, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 5.2393, 95% CI 2-sided [-0.2058 to 10.6845], Standard Error of Mean 2.7396
Statistical Analysis 7: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; Day 113 : Adjusted mean difference and 2-sided 95% confidence interval were derived from the MMRM model with fixed effects for treatment, visit, baseline value, treatment by visit interaction, and baseline by visit interaction; Test type: Superiority or Other; p = 0.185, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 2.1827, 95% CI 2-sided [-2.6334 to 6.9988], Standard Error of Mean 2.4251
Statistical Analysis 8: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.195, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 2.1376, 95% CI 2-sided [-2.7718 to 7.0469], Standard Error of Mean 2.4716
Statistical Analysis 9: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.450, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 0.3113, 95% CI 2-sided [-4.6358 to 5.2584], Standard Error of Mean 2.4909
Statistical Analysis 10: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.397, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 0.6078, 95% CI 2-sided [-4.0274 to 5.2431], Standard Error of Mean 2.3322
Statistical Analysis 11: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.008, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 5.7096, 95% CI 2-sided [1.0659 to 10.3532], Standard Error of Mean 2.3367
Statistical Analysis 12: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 12]; Test type: Superiority or Other; p = 0.147, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 2.4558, 95% CI 2-sided [-2.1608 to 7.0724], Standard Error of Mean 2.3230

17. Secondary Outcome: Lipoprotein (a) (Lp[a])
Description: Lp(a) is a lipoprotein subclass which consists of an LDL-like particle and the specific apolipoprotein(a). Fasting was required at least 10 hours before blood sample collection. Baseline was defined as the mean of the last two non-missing measurements collected prior to the first dose of study treatment. Both measurements must be within 10 days prior to the first dose of study treatment; if only one measurement was available 10 days prior to the first dose of study treatment, then that measurement served as the baseline value.
Time Frame: Baseline, Day 5, 8, 15, 22, 29, 36, 43, 50, 57, 71, 85, 99, 106, 113, 127, 141, 155, 169
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 26 | 22 | 25 | 25 | 24 | 23
mg/dL
  Baseline | 18.452 (13.1792) | 20.998 (17.2111) | 18.840 (16.7289) | 19.265 (14.3646) | 19.468 (18.4181) | 14.080 (11.9369) | 15.458 (12.6296) | 13.400 (9.0719) | 16.239 (10.1883)
  Day 5: number analyzed (Participants) | 25 | 23 | 23 | 26 | 22 | 25 | 25 | 24 | 22
  Day 5 | 16.224 (13.4935) | 18.348 (17.7316) | 16.204 (16.6072) | 18.523 (15.2512) | 20.450 (18.8904) | 12.464 (10.5751) | 14.580 (12.2541) | 11.783 (9.3506) | 15.859 (10.9932)
  Day 8: number analyzed (Participants) | 25 | 24 | 24 | 25 | 21 | 25 | 24 | 22 | 23
  Day 8 | 14.892 (13.2944) | 15.333 (18.3499) | 14.167 (15.5022) | 19.184 (14.7461) | 17.243 (15.7353) | 12.000 (11.8358) | 12.617 (10.4189) | 12.768 (8.9168) | 16.443 (12.1793)
  Day 15 | 14.208 (12.9280) | 14.129 (17.8567) | 11.392 (14.1251) | 19.258 (16.0484) | 18.982 (20.4348) | 10.140 (10.0017) | 12.548 (10.9860) | 9.996 (8.1113) | 16.443 (11.4594)
  Day 22: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 22 | 12.628 (12.4393) | 12.446 (16.1397) | 10.765 (13.3504) | 18.785 (16.0604) | 17.800 (18.6499) | 10.936 (10.1920) | 11.583 (11.3914) | 8.800 (7.1835) | 16.026 (11.0080)
  Day 29: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 25 | 25 | 24 | 22
  Day 29 | 12.832 (12.3874) | 13.379 (16.2405) | 10.552 (12.7986) | 18.304 (15.6050) | 17.873 (18.0678) | 10.424 (10.6085) | 10.888 (9.8450) | 9.312 (7.3675) | 17.423 (11.1746)
  Day 36: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 36 | 11.152 (11.9088) | 12.833 (16.0418) | 10.409 (12.7145) | 17.046 (14.4893) | 18.050 (19.5448) | 9.484 (10.6692) | 10.329 (9.7943) | 8.067 (6.7186) | 15.843 (10.8050)
  Day 43 | 11.648 (12.2798) | 12.525 (16.1360) | 9.633 (12.4360) | 16.912 (14.1356) | 17.214 (18.6825) | 9.380 (9.6416) | 9.944 (9.7431) | 8.821 (7.6426) | 15.961 (10.3890)
  Day 50: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Day 50 | 10.344 (11.3684) | 11.675 (14.8818) | 9.039 (12.0250) | 16.835 (14.2068) | 17.314 (19.6439) | 10.040 (10.4835) | 10.191 (9.2630) | 7.621 (6.5659) | 15.078 (9.7608)
  Day 57: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 57 | 10.708 (10.3883) | 10.871 (13.5224) | 8.578 (11.2275) | 15.892 (14.0990) | 17.573 (21.9401) | 9.392 (10.2457) | 9.487 (8.2801) | 6.858 (6.2894) | 14.313 (9.3930)
  Day 71: number analyzed (Participants) | 24 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 71 | 11.358 (12.3793) | 11.354 (14.0492) | 9.009 (11.7733) | 16.542 (13.5029) | 16.991 (20.0151) | 9.248 (11.4972) | 9.529 (8.6412) | 6.979 (6.5414) | 13.500 (9.4333)
  Day 85: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Day 85 | 10.960 (11.6806) | 10.879 (14.1289) | 9.239 (11.1448) | 16.519 (14.5691) | 17.609 (19.7001) | 8.808 (10.3417) | 9.261 (7.6804) | 6.637 (5.6695) | 12.726 (8.9598)
  Day 99: number analyzed (Participants) | 25 | 24 | 22 | 25 | 22 | 25 | 24 | 24 | 23
  Day 99 | 12.232 (12.5326) | 11.837 (15.6082) | 8.855 (13.9399) | 15.764 (14.4527) | 16.868 (19.6709) | 7.940 (9.6343) | 8.537 (7.6094) | 6.792 (5.6212) | 13.691 (9.5937)
  Day 106: number analyzed (Participants) | 25 | 24 | 22 | 25 | 22 | 25 | 23 | 24 | 23
  Day 106 | 10.756 (11.7377) | 11.079 (14.2590) | 9.123 (14.1064) | 15.396 (12.8944) | 16.682 (18.8434) | 8.608 (9.5662) | 8.296 (7.3410) | 6.858 (6.1058) | 12.800 (8.9601)
  Day 113: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 23 | 23
  Day 113 | 12.108 (12.3479) | 11.183 (14.5312) | 9.565 (14.0691) | 14.492 (12.9060) | 16.814 (17.8976) | 8.020 (9.0412) | 8.287 (7.6439) | 6.787 (5.8743) | 12.913 (9.7212)
  Day 127: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 25 | 23 | 24 | 23
  Day 127 | 15.476 (14.6308) | 15.112 (16.5781) | 11.961 (15.6073) | 15.500 (13.0255) | 16.618 (19.1791) | 9.864 (10.2016) | 10.543 (9.2205) | 7.642 (6.9977) | 13.596 (9.3340)
  Day 141: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 24 | 23
  Day 141 | 16.842 (15.6809) | 17.329 (18.9837) | 14.422 (17.3620) | 15.828 (13.7114) | 17.236 (18.8525) | 10.100 (10.9325) | 11.996 (10.0494) | 8.442 (6.7945) | 13.139 (9.2951)
  Day 155: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 23 | 23 | 24 | 23
  Day 155 | 17.264 (15.4506) | 17.483 (19.9385) | 16.052 (16.9174) | 16.004 (13.7418) | 17.382 (19.8297) | 10.204 (11.2720) | 13.465 (10.8114) | 9.600 (7.5028) | 13.183 (9.1710)
  Day 169: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 24 | 23 | 23 | 22
  Day 169 | 17.824 (15.1879) | 17.404 (18.0405) | 16.635 (17.8211) | 15.384 (13.7150) | 17.059 (20.8409) | 11.271 (11.4561) | 13.613 (11.5074) | 10.626 (8.0902) | 14.741 (10.3647)

18. Secondary Outcome: Change From Baseline in Lipoprotein (a) (Lp[a]) at Day 85 and Day 113
Description: Lp(a) is a lipoprotein subclass which consists of an LDL-like particle and the specific apolipoprotein(a). Fasting was required at least 10 hours before blood sample collection. Baseline was defined as the mean of the last two non-missing measurements collected prior to the first dose of study treatment. Both measurements must be within 10 days prior to the first dose of study treatment; if only one measurement was available 10 days prior to the first dose of study treatment, then that measurement served as the baseline value. Change from baseline = observed value minus baseline value.
Time Frame: Baseline, Day 85, 113
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 26 | 22 | 25 | 25 | 24 | 23
mg/dL
  Change at Day 85: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Change at Day 85 | -7.492 (5.1400) | -10.119 (5.4374) | -10.239 (8.2471) | -2.746 (3.1292) | -1.859 (3.0759) | -5.272 (5.1528) | -7.100 (5.9402) | -6.763 (5.3474) | -3.513 (3.6550)
  Change at Day 113: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 23 | 23
  Change at Day 113 | -6.815 (4.6182) | -9.815 (5.0568) | -9.913 (6.6763) | -3.574 (4.0251) | -2.655 (3.1725) | -6.060 (4.5477) | -8.074 (6.0886) | -7.098 (4.5025) | -3.326 (3.4975)
Statistical Analysis 1: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -4.9203, 95% CI 2-sided [-7.5504 to -2.2901], Standard Error of Mean 1.3242
Statistical Analysis 2: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -7.1983, 95% CI 2-sided [-9.8718 to -4.5249], Standard Error of Mean 1.3462
Statistical Analysis 3: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -7.3118, 95% CI 2-sided [-9.9935 to -4.6301], Standard Error of Mean 1.3505
Statistical Analysis 4: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -3.0629, 95% CI 2-sided [-5.1132 to -1.0125], Standard Error of Mean 1.0320
Statistical Analysis 5: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -3.6209, 95% CI 2-sided [-5.6804 to -1.5614], Standard Error of Mean 1.0367
Statistical Analysis 6: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -4.1778, 95% CI 2-sided [-6.2184 to -2.1372], Standard Error of Mean 1.0269
Statistical Analysis 7: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.006, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -3.2914, 95% CI 2-sided [-5.8649 to -0.7178], Standard Error of Mean 1.2954
Statistical Analysis 8: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -6.3569, 95% CI 2-sided [-8.9706 to -3.7432], Standard Error of Mean 1.3157
Statistical Analysis 9: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -6.3962, 95% CI 2-sided [-9.0247 to -3.7677], Standard Error of Mean 1.3233
Statistical Analysis 10: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -3.9228, 95% CI 2-sided [-5.7506 to -2.0950], Standard Error of Mean 0.9199
Statistical Analysis 11: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -4.7094, 95% CI 2-sided [-6.5459 to -2.8729], Standard Error of Mean 0.9244
Statistical Analysis 12: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 12]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -4.4374, 95% CI 2-sided [-6.2630 to -2.6118], Standard Error of Mean 0.9187

19. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a) (Lp[a]) at Day 85 and Day 113
Description: Lp(a) is a lipoprotein subclass which consists of an LDL-like particle and the specific apolipoprotein(a). Fasting was required at least 10 hours before blood sample collection. Baseline was defined as the mean of the last two non-missing measurements collected prior to the first dose of study treatment. Both measurements must be within 10 days prior to the first dose of study treatment; if only one measurement was available 10 days prior to the first dose of study treatment, then that measurement served as the baseline value. Percent change from baseline = ([observed value divided by baseline value] minus 1) multiplied by 100.
Time Frame: Baseline, Day 85, 113
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 26 | 22 | 25 | 25 | 24 | 23
percent change
  Change at Day 85: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Change at Day 85 | -47.11 (20.802) | -58.53 (22.181) | -46.51 (63.192) | -19.37 (25.160) | -15.22 (23.532) | -37.85 (27.223) | -37.29 (24.552) | -43.37 (39.755) | -18.40 (30.139)
  Change at Day 113: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 23 | 23
  Change at Day 113 | -42.30 (19.223) | -57.94 (22.317) | -59.42 (21.689) | -24.35 (21.348) | -18.64 (18.300) | -45.26 (22.490) | -47.60 (19.448) | -49.77 (25.417) | -15.89 (36.642)
Statistical Analysis 1: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -27.4492, 95% CI 2-sided [-47.7872 to -7.1112], Standard Error of Mean 10.2401
Statistical Analysis 2: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -40.5908, 95% CI 2-sided [-61.3577 to -19.8240], Standard Error of Mean 10.4568
Statistical Analysis 3: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.006, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -27.1630, 95% CI 2-sided [-48.0927 to -6.2332], Standard Error of Mean 10.5402
Statistical Analysis 4: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -24.1677, 95% CI 2-sided [-41.8023 to -6.5332], Standard Error of Mean 8.8755
Statistical Analysis 5: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.017, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -19.2255, 95% CI 2-sided [-36.9471 to -1.5038], Standard Error of Mean 8.9203
Statistical Analysis 6: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -26.5155, 95% CI 2-sided [-44.0795 to -8.9515], Standard Error of Mean 8.8387
Statistical Analysis 7: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -18.3898, 95% CI 2-sided [-28.6698 to -8.1097], Standard Error of Mean 5.1768
Statistical Analysis 8: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -36.7882, 95% CI 2-sided [-47.2423 to -26.3341], Standard Error of Mean 5.2640
Statistical Analysis 9: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -36.8453, 95% CI 2-sided [-47.3864 to -26.3041], Standard Error of Mean 5.3084
Statistical Analysis 10: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -32.9411, 95% CI 2-sided [-48.5748 to -17.3075], Standard Error of Mean 7.8656
Statistical Analysis 11: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -31.3176, 95% CI 2-sided [-47.0238 to -15.6114], Standard Error of Mean 7.9032
Statistical Analysis 12: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 12]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -32.8470, 95% CI 2-sided [-48.4650 to -17.2289], Standard Error of Mean 7.8576

20. Secondary Outcome: High Density Lipoprotein- Cholesterol (HDL-C)
Description: HDL-C is cholesterol in the bloodstream that is carried by high density lipoprotein. Fasting was required at least 10 hours before blood sample collection. Baseline was defined as the mean of the last two non-missing measurements collected prior to the first dose of study treatment. Both measurements must be within 10 days prior to the first dose of study treatment; if only one measurement was available 10 days prior to the first dose of study treatment, then that measurement served as the baseline value.
Time Frame: Baseline, Day 5, 8, 15, 22, 29, 36, 43, 50, 57, 71, 85, 99, 106, 113, 127, 141, 155, 169
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 26 | 22 | 25 | 25 | 24 | 23
mg/dL
  Baseline | 54.58 (9.048) | 54.75 (11.789) | 57.00 (12.858) | 58.54 (14.683) | 56.98 (9.607) | 57.22 (14.146) | 60.40 (13.228) | 62.02 (21.455) | 60.87 (10.606)
  Day 5: number analyzed (Participants) | 25 | 23 | 23 | 26 | 22 | 25 | 25 | 24 | 22
  Day 5 | 55.68 (11.131) | 57.04 (12.532) | 58.43 (13.480) | 58.19 (14.403) | 57.00 (9.866) | 57.20 (15.785) | 60.32 (13.643) | 62.08 (21.354) | 59.73 (11.344)
  Day 8: number analyzed (Participants) | 25 | 24 | 24 | 25 | 21 | 25 | 24 | 22 | 23
  Day 8 | 56.48 (11.266) | 58.38 (12.700) | 60.33 (13.017) | 60.52 (14.234) | 58.67 (10.136) | 59.60 (15.729) | 61.33 (14.230) | 64.00 (23.420) | 60.57 (11.289)
  Day 15 | 58.52 (8.637) | 59.96 (11.925) | 62.79 (15.562) | 59.35 (15.179) | 60.23 (12.208) | 60.24 (16.048) | 62.32 (15.513) | 66.58 (22.085) | 60.30 (11.117)
  Day 22: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 22 | 59.36 (11.158) | 60.08 (12.176) | 64.52 (14.585) | 58.08 (12.743) | 60.05 (10.017) | 60.92 (16.253) | 63.92 (13.529) | 65.38 (17.358) | 61.48 (11.233)
  Day 29: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 25 | 25 | 24 | 22
  Day 29 | 59.96 (10.486) | 61.75 (13.553) | 63.83 (15.948) | 57.96 (13.192) | 59.00 (9.587) | 60.84 (16.222) | 62.52 (15.196) | 67.96 (20.412) | 64.14 (9.896)
  Day 36: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 36 | 57.92 (10.622) | 60.50 (13.112) | 62.39 (14.151) | 57.62 (13.518) | 58.23 (10.314) | 59.76 (14.521) | 65.25 (14.411) | 65.21 (19.489) | 59.91 (10.833)
  Day 43 | 59.76 (8.724) | 62.21 (13.266) | 62.29 (15.415) | 57.31 (13.936) | 58.82 (10.450) | 59.36 (14.950) | 63.64 (15.435) | 65.17 (18.846) | 59.74 (10.558)
  Day 50: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Day 50 | 60.12 (10.248) | 60.04 (12.185) | 62.09 (14.058) | 57.81 (14.525) | 58.55 (10.835) | 59.40 (14.955) | 64.91 (13.651) | 65.21 (19.669) | 59.39 (10.586)
  Day 57: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 57 | 58.40 (8.221) | 58.83 (13.830) | 60.35 (13.231) | 54.88 (12.745) | 57.45 (10.804) | 57.16 (12.589) | 61.92 (14.374) | 62.63 (20.549) | 56.61 (10.782)
  Day 71: number analyzed (Participants) | 24 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 71 | 60.29 (9.438) | 62.96 (14.0492) | 64.83 (16.854) | 56.85 (12.069) | 58.00 (9.798) | 59.16 (13.539) | 63.92 (14.185) | 66.29 (20.354) | 57.78 (9.662)
  Day 85: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Day 85 | 58.24 (9.926) | 59.54 (12.827) | 59.70 (11.315) | 53.96 (12.981) | 59.77 (10.438) | 55.04 (13.421) | 63.09 (13.211) | 62.00 (17.619) | 56.35 (10.075)
  Day 99: number analyzed (Participants) | 25 | 24 | 22 | 25 | 22 | 25 | 24 | 24 | 23
  Day 99 | 62.68 (11.926) | 62.54 (13.462) | 62.32 (14.496) | 59.92 (12.812) | 60.36 (10.472) | 60.00 (13.051) | 64.54 (15.453) | 64.63 (18.946) | 59.30 (12.430)
  Day 106: number analyzed (Participants) | 25 | 24 | 22 | 25 | 22 | 25 | 23 | 24 | 23
  Day 106 | 62.36 (11.489) | 63.25 (15.118) | 64.41 (13.355) | 58.28 (12.651) | 59.45 (10.117) | 60.08 (15.231) | 64.39 (15.718) | 65.17 (18.897) | 58.30 (11.703)
  Day 113: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 23 | 23
  Day 113 | 58.13 (11.395) | 61.04 (14.245) | 59.39 (12.565) | 55.28 (13.145) | 60.32 (10.049) | 57.92 (14.617) | 63.00 (14.331) | 61.83 (18.218) | 56.17 (10.421)
  Day 127: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 25 | 23 | 24 | 23
  Day 127 | 59.16 (12.212) | 59.46 (13.552) | 62.78 (14.013) | 60.72 (15.118) | 57.82 (9.272) | 58.56 (13.818) | 63.61 (16.160) | 63.88 (19.161) | 58.00 (10.838)
  Day 141: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 24 | 23
  Day 141 | 60.58 (11.960) | 60.63 (13.682) | 64.26 (14.530) | 60.96 (15.970) | 59.09 (10.766) | 59.40 (16.081) | 63.26 (14.229) | 64.00 (20.167) | 62.39 (14.138)
  Day 155: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 23 | 23 | 24 | 23
  Day 155 | 58.72 (10.620) | 59.00 (14.341) | 61.96 (14.455) | 59.48 (14.535) | 59.45 (9.179) | 59.04 (16.425) | 63.00 (15.021) | 63.67 (20.550) | 61.87 (13.602)
  Day 169: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 24 | 23 | 23 | 22
  Day 169 | 57.48 (11.794) | 59.04 (12.726) | 62.48 (14.441) | 61.88 (15.078) | 60.50 (11.827) | 60.29 (16.206) | 62.04 (15.155) | 65.00 (24.355) | 65.05 (13.584)

21. Secondary Outcome: Change From Baseline in High Density Lipoprotein- Cholesterol (HDL-C) at Day 85 and Day 113
Description: HDL-C is cholesterol in the bloodstream that is carried by high density lipoprotein. Fasting was required at least 10 hours before blood sample collection. Baseline was defined as the mean of the last two non-missing measurements collected prior to the first dose of study treatment. Both measurements must be within 10 days prior to the first dose of study treatment; if only one measurement was available 10 days prior to the first dose of study treatment, then that measurement served as the baseline value. Change from baseline = observed value minus baseline value.
Time Frame: Baseline, Day 85, 113
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 26 | 22 | 25 | 25 | 24 | 23
mg/dL
  Change at Day 85: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Change at Day 85 | 3.66 (6.216) | 4.79 (5.568) | 2.63 (5.394) | -4.58 (4.573) | 2.80 (6.223) | -2.18 (6.065) | 1.46 (7.408) | -0.02 (7.575) | -4.52 (5.191)
  Change at Day 113: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 23 | 23
  Change at Day 113 | 3.90 (6.437) | 6.29 (7.003) | 2.33 (8.053) | -3.28 (7.264) | 3.34 (5.702) | 0.70 (6.489) | 1.37 (7.799) | -0.63 (6.995) | -4.70 (5.045)
Statistical Analysis 1: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 7.663, 95% CI 2-sided [4.820 to 10.506], Standard Error of Mean 1.431
Statistical Analysis 2: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 9.290, 95% CI 2-sided [6.389 to 12.190], Standard Error of Mean 1.460
Statistical Analysis 3: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 7.255, 95% CI 2-sided [4.336 to 10.175], Standard Error of Mean 1.470
Statistical Analysis 4: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.110, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 2.228, 95% CI 2-sided [-1.361 to 5.818], Standard Error of Mean 1.806
Statistical Analysis 5: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 5.578, 95% CI 2-sided [1.972 to 9.185], Standard Error of Mean 1.815
Statistical Analysis 6: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 4.712, 95% CI 2-sided [1.156 to 8.268], Standard Error of Mean 1.789
Statistical Analysis 7: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 5.888, 95% CI 2-sided [1.844 to 9.932], Standard Error of Mean 2.035
Statistical Analysis 8: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 9.251, 95% CI 2-sided [5.153 to 13.349], Standard Error of Mean 2.062
Statistical Analysis 9: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.006, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 5.264, 95% CI 2-sided [1.147 to 9.380], Standard Error of Mean 2.072
Statistical Analysis 10: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 5.065, 95% CI 2-sided [1.402 to 8.728], Standard Error of Mean 1.843
Statistical Analysis 11: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 5.096, 95% CI 2-sided [1.413 to 8.780], Standard Error of Mean 1.853
Statistical Analysis 12: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 12]; Test type: Superiority or Other; p = 0.011, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 4.301, 95% CI 2-sided [0.658 to 7.943], Standard Error of Mean 1.832

22. Secondary Outcome: Percent Change From Baseline in High Density Lipoprotein- Cholesterol (HDL-C) at Day 85 and Day 113
Description: HDL-C is cholesterol in the bloodstream that is carried by high density lipoprotein. Fasting was required at least 10 hours before blood sample collection. Baseline was defined as the mean of the last two non-missing measurements collected prior to the first dose of study treatment. Both measurements must be within 10 days prior to the first dose of study treatment; if only one measurement was available 10 days prior to the first dose of study treatment, then that measurement served as the baseline value. Percent change from baseline = ([observed value divided by baseline value] minus 1) multiplied by 100.
Time Frame: Baseline, Day 85, 113
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 26 | 22 | 25 | 25 | 24 | 23
percent change
  Change at Day 85: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Change at Day 85 | 7.26 (10.914) | 9.46 (11.132) | 5.86 (9.988) | -7.31 (7.254) | 5.42 (10.501) | -3.10 (10.471) | 2.93 (11.259) | 2.35 (12.101) | -7.16 (8.271)
  Change at Day 113: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 23 | 23
  Change at Day 113 | 7.39 (11.623) | 11.97 (13.385) | 5.27 (12.612) | -4.83 (9.919) | 6.31 (9.989) | 1.86 (11.617) | 2.35 (10.959) | 1.05 (10.017) | -7.53 (7.966)
Statistical Analysis 1: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 13.389, 95% CI 2-sided [8.373 to 18.405], Standard Error of Mean 2.525
Statistical Analysis 2: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 16.546, 95% CI 2-sided [11.430 to 21.663], Standard Error of Mean 2.576
Statistical Analysis 3: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 13.288, 95% CI 2-sided [8.137 to 18.438], Standard Error of Mean 2.593
Statistical Analysis 4: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.081, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 4.112, 95% CI 2-sided [-1.671 to 9.895], Standard Error of Mean 2.909
Statistical Analysis 5: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 9.560, 95% CI 2-sided [3.743 to 15.377], Standard Error of Mean 2.927
Statistical Analysis 6: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 9.826, 95% CI 2-sided [4.103 to 15.548], Standard Error of Mean 2.878
Statistical Analysis 7: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 10.004, 95% CI 2-sided [3.395 to 16.612], Standard Error of Mean 3.326
Statistical Analysis 8: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 16.252, 95% CI 2-sided [9.560 to 22.943], Standard Error of Mean 3.367
Statistical Analysis 9: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 9.571, 95% CI 2-sided [2.847 to 16.295], Standard Error of Mean 3.384
Statistical Analysis 10: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 9.029, 95% CI 2-sided [3.348 to 14.710], Standard Error of Mean 2.858
Statistical Analysis 11: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 8.543, 95% CI 2-sided [2.827 to 14.260], Standard Error of Mean 2.876
Statistical Analysis 12: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 12]; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 8.898, 95% CI 2-sided [3.252 to 14.544], Standard Error of Mean 2.840

23. Secondary Outcome: Very Low Density Lipoprotein-Cholesterol (VLDL-C)
Description: VLDL is a type of lipoprotein made by the liver and one of the five major groups of lipoproteins, that enable fats and cholesterol to move within the water-based solution of the bloodstream. Fasting was required at least 10 hours before blood sample collection. Baseline was defined as the mean of the last two non-missing measurements collected prior to the first dose of study treatment. Both measurements must be within 10 days prior to the first dose of study treatment; if only one measurement was available 10 days prior to the first dose of study treatment, then that measurement served as the baseline value.
Time Frame: Baseline, Day 5, 8, 15, 22, 29, 36, 43, 50, 57, 71, 85, 99, 106, 113, 127, 141, 155, 169
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 26 | 22 | 25 | 25 | 24 | 23
mg/dL
  Baseline | 19.92 (9.312) | 23.79 (11.286) | 20.92 (7.651) | 21.42 (6.858) | 22.48 (7.869) | 17.44 (7.509) | 17.66 (9.090) | 16.63 (6.273) | 17.50 (8.549)
  Day 5: number analyzed (Participants) | 25 | 23 | 23 | 26 | 22 | 25 | 25 | 24 | 22
  Day 5 | 21.36 (9.999) | 19.70 (8.249) | 17.22 (5.977) | 23.85 (10.657) | 21.95 (8.249) | 19.80 (11.927) | 16.08 (8.356) | 18.00 (10.065) | 20.68 (10.035)
  Day 8: number analyzed (Participants) | 25 | 24 | 24 | 25 | 21 | 25 | 24 | 22 | 23
  Day 8 | 19.64 (13.073) | 18.00 (6.574) | 15.58 (6.192) | 21.72 (10.577) | 20.29 (7.100) | 18.64 (9.995) | 16.25 (6.661) | 18.95 (9.810) | 22.48 (13.737)
  Day 15 | 17.20 (8.921) | 20.42 (9.930) | 16.50 (9.869) | 23.04 (9.035) | 22.68 (9.712) | 18.52 (9.265) | 16.28 (8.735) | 16.25 (10.605) | 20.43 (10.612)
  Day 22: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 22 | 17.04 (6.761) | 19.04 (7.410) | 14.65 (6.786) | 21.65 (7.573) | 21.59 (7.866) | 17.20 (7.984) | 16.42 (6.580) | 17.17 (14.199) | 18.13 (9.416)
  Day 29: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 25 | 25 | 24 | 22
  Day 29 | 15.76 (7.253) | 19.88 (9.967) | 15.39 (4.717) | 21.88 (9.523) | 22.73 (10.552) | 17.00 (7.746) | 19.68 (16.106) | 13.04 (6.753) | 19.00 (8.258)
  Day 36: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 36 | 18.96 (9.361) | 15.33 (4.984) | 14.04 (5.842) | 21.92 (9.587) | 21.59 (9.169) | 17.28 (6.901) | 16.46 (6.129) | 15.50 (5.905) | 24.22 (17.231)
  Day 43 | 16.56 (6.246) | 21.33 (13.770) | 18.04 (10.813) | 23.65 (12.547) | 20.95 (7.712) | 20.00 (7.708) | 18.12 (7.316) | 16.96 (6.734) | 22.78 (11.631)
  Day 50: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Day 50 | 16.36 (9.269) | 17.67 (6.787) | 14.39 (6.966) | 21.69 (11.235) | 19.23 (6.718) | 17.48 (8.186) | 17.04 (7.151) | 15.54 (7.818) | 22.26 (13.685)
  Day 57: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 57 | 14.36 (6.034) | 17.46 (8.939) | 13.87 (4.674) | 20.88 (7.957) | 21.55 (5.878) | 15.44 (5.108) | 16.83 (12.437) | 13.54 (4.222) | 20.13 (10.092)
  Day 71: number analyzed (Participants) | 24 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 71 | 15.92 (7.064) | 17.50 (9.212) | 13.83 (3.950) | 21.77 (9.868) | 20.82 (8.151) | 19.04 (6.846) | 16.79 (6.840) | 14.63 (6.337) | 22.61 (9.014)
  Day 85: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Day 85 | 14.24 (6.247) | 17.63 (8.816) | 14.04 (6.745) | 22.58 (7.991) | 19.77 (5.936) | 16.68 (7.040) | 14.09 (6.735) | 14.04 (4.639) | 16.43 (8.877)
  Day 99: number analyzed (Participants) | 25 | 24 | 22 | 25 | 22 | 25 | 24 | 24 | 23
  Day 99 | 16.20 (6.371) | 18.04 (10.378) | 18.68 (17.700) | 21.72 (11.085) | 20.14 (7.298) | 17.84 (6.756) | 16.46 (9.514) | 16.21 (8.490) | 21.13 (8.981)
  Day 106: number analyzed (Participants) | 25 | 24 | 22 | 25 | 22 | 25 | 23 | 24 | 23
  Day 106 | 14.44 (6.545) | 15.96 (6.328) | 14.59 (5.981) | 19.32 (7.330) | 18.64 (6.499) | 17.76 (7.573) | 16.09 (5.672) | 13.13 (5.788) | 20.00 (9.376)
  Day 113: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 23 | 23
  Day 113 | 15.83 (8.726) | 16.54 (7.863) | 15.26 (5.056) | 21.88 (14.701) | 18.50 (7.951) | 15.92 (8.246) | 15.96 (8.466) | 13.87 (6.107) | 19.39 (8.322)
  Day 127: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 25 | 23 | 24 | 23
  Day 127 | 20.48 (11.594) | 23.21 (14.231) | 16.61 (7.686) | 19.32 (9.534) | 21.59 (7.992) | 19.72 (8.091) | 17.91 (11.445) | 17.38 (12.631) | 21.61 (13.121)
  Day 141: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 24 | 23
  Day 141 | 18.13 (7.279) | 22.25 (15.109) | 17.39 (5.007) | 19.16 (9.573) | 23.68 (9.564) | 19.52 (10.627) | 17.61 (7.518) | 18.54 (9.913) | 20.09 (9.409)
  Day 155: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 23 | 23 | 24 | 23
  Day 155 | 17.00 (3.905) | 22.21 (11.858) | 16.52 (7.141) | 20.56 (9.319) | 21.41 (7.028) | 19.30 (9.632) | 16.17 (8.144) | 18.92 (10.738) | 18.57 (9.110)
  Day 169: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 24 | 23 | 23 | 22
  Day 169 | 18.88 (7.732) | 21.42 (7.442) | 17.30 (6.292) | 19.60 (7.286) | 24.55 (11.931) | 19.13 (8.644) | 23.00 (23.279) | 18.00 (10.167) | 19.68 (8.306)

24. Secondary Outcome: Change From Baseline in Very Low Density Lipoprotein-Cholesterol (VLDL-C) at Day 85 and Day 113
Description: VLDL is a type of lipoprotein made by the liver and one of the five major groups of lipoproteins, that enable fats and cholesterol to move within the water-based solution of the bloodstream. Fasting was required at least 10 hours before blood sample collection. Baseline was defined as the mean of the last two non-missing measurements collected prior to the first dose of study treatment. Both measurements must be within 10 days prior to the first dose of study treatment; if only one measurement was available 10 days prior to the first dose of study treatment, then that measurement served as the baseline value. Change from baseline = observed value minus baseline value.
Time Frame: Baseline, Day 85, 113
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 26 | 22 | 25 | 25 | 24 | 23
mg/dL
  Change at Day 85: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Change at Day 85 | -5.68 (6.973) | -6.17 (7.171) | -6.57 (6.726) | 1.15 (4.841) | -2.70 (7.069) | -0.76 (5.114) | -2.63 (9.497) | -2.58 (7.290) | -1.07 (4.989)
  Change at Day 113: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 23 | 23
  Change at Day 113 | -4.29 (8.538) | -7.25 (9.067) | -5.35 (6.619) | 0.34 (10.957) | -3.98 (8.873) | -1.52 (5.771) | -0.76 (9.276) | -2.98 (6.998) | 1.89 (5.762)
Statistical Analysis 1: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -7.462, 95% CI 2-sided [-10.311 to -4.614], Standard Error of Mean 1.434
Statistical Analysis 2: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -6.693, 95% CI 2-sided [-9.610 to -3.776], Standard Error of Mean 1.469
Statistical Analysis 3: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -8.755, 95% CI 2-sided [-11.692 to -5.817], Standard Error of Mean 1.479
Statistical Analysis 4: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.484, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -0.072, 95% CI 2-sided [-3.596 to 3.451], Standard Error of Mean 1.773
Statistical Analysis 5: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.173, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -1.701, 95% CI 2-sided [-5.264 to 1.862], Standard Error of Mean 1.793
Statistical Analysis 6: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.135, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -1.953, 95% CI 2-sided [-5.452 to 1.546], Standard Error of Mean 1.761
Statistical Analysis 7: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.034, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -4.447, 95% CI 2-sided [-9.230 to 0.335], Standard Error of Mean 2.406
Statistical Analysis 8: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -6.764, 95% CI 2-sided [-11.617 to -1.910], Standard Error of Mean 2.442
Statistical Analysis 9: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.009, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -5.951, 95% CI 2-sided [-10.836 to -1.066], Standard Error of Mean 2.458
Statistical Analysis 10: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.056, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -3.070, 95% CI 2-sided [-6.876 to 0.736], Standard Error of Mean 1.915
Statistical Analysis 11: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.095, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -2.557, 95% CI 2-sided [-6.408 to 1.293], Standard Error of Mean 1.937
Statistical Analysis 12: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 12]; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -5.271, 95% CI 2-sided [-9.074 to -1.469], Standard Error of Mean 1.913

25. Secondary Outcome: Percent Change From Baseline in Very Low Density Lipoprotein-Cholesterol (VLDL-C) at Day 85 and Day 113
Description: VLDL is a type of lipoprotein made by the liver and one of the five major groups of lipoproteins, that enable fats and cholesterol to move within the water-based solution of the bloodstream. Fasting was required at least 10 hours before blood sample collection. Baseline was defined as the mean of the last two non-missing measurements collected prior to the first dose of study treatment. Both measurements must be within 10 days prior to the first dose of study treatment; if only one measurement was available 10 days prior to the first dose of study treatment, then that measurement served as the baseline value. Percent change from baseline = ([observed value divided by baseline value] minus 1) multiplied by 100.
Time Frame: Baseline, Day 85, 113
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 26 | 22 | 25 | 25 | 24 | 23
percent change
  Change at Day 85: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 24 | 23 | 24 | 23
  Change at Day 85 | -23.42 (30.458) | -22.99 (25.647) | -28.96 (25.281) | 7.08 (26.054) | -6.48 (27.276) | -7.61 (23.163) | 5.66 (76.931) | -3.54 (45.821) | -3.63 (39.826)
  Change at Day 113: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 24 | 23 | 23 | 23
  Change at Day 113 | -17.23 (35.083) | -26.62 (28.464) | -19.28 (33.794) | -1.89 (43.239) | -10.80 (38.288) | -9.72 (29.006) | 10.72 (65.297) | -10.36 (36.732) | 18.73 (48.065)
Statistical Analysis 1: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -31.880, 95% CI 2-sided [-45.925 to -17.836], Standard Error of Mean 7.071
Statistical Analysis 2: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -29.187, 95% CI 2-sided [-43.571 to -14.803], Standard Error of Mean 7.242
Statistical Analysis 3: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -39.657, 95% CI 2-sided [-54.136 to -25.178], Standard Error of Mean 7.290
Statistical Analysis 4: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.366, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -4.681, 95% CI 2-sided [-31.713 to 22.350], Standard Error of Mean 13.601
Statistical Analysis 5: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.773, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 10.227, 95% CI 2-sided [-16.774 to 37.228], Standard Error of Mean 13.586
Statistical Analysis 6: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.422, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -2.646, 95% CI 2-sided [-29.206 to 23.915], Standard Error of Mean 13.362
Statistical Analysis 7: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.107, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -12.911, 95% CI 2-sided [-33.411 to 7.589], Standard Error of Mean 10.309
Statistical Analysis 8: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.015, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -23.119, 95% CI 2-sided [-43.923 to -2.315], Standard Error of Mean 10.461
Statistical Analysis 9: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.054, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -17.159, 95% CI 2-sided [-38.108 to 3.789], Standard Error of Mean 10.535
Statistical Analysis 10: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.029, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -24.416, 95% CI 2-sided [-49.696 to 0.865], Standard Error of Mean 12.718
Statistical Analysis 11: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.311, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -6.287, 95% CI 2-sided [-31.541 to 18.968], Standard Error of Mean 12.705
Statistical Analysis 12: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 12]; Test type: Superiority or Other; p = 0.006, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -32.443, 95% CI 2-sided [-57.400 to -7.485], Standard Error of Mean 12.555

26. Secondary Outcome: Triglyceride (TG)
Description: Triglycerides are a type of fat circulating in the blood and account for the majority of the fats circulating in the blood. Fasting was required at least 10 hours before blood sample collection. Baseline was defined as the mean of the last two non-missing measurements collected prior to the first dose of study treatment. Both measurements must be within 10 days prior to the first dose of study treatment; if only one measurement was available 10 days prior to the first dose of study treatment, then that measurement served as the baseline value.
Time Frame: Baseline, Day 5, 8, 15, 22, 29, 36, 43, 50, 57, 71, 85, 99, 106, 113, 127, 141, 155, 169
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 26 | 22 | 25 | 25 | 24 | 23
mg/dL
  Baseline | 121.04 (56.152) | 158.21 (71.477) | 127.65 (59.878) | 140.23 (51.283) | 152.59 (50.105) | 122.40 (50.578) | 124.40 (59.717) | 111.58 (42.354) | 130.39 (49.826)
  Day 5: number analyzed (Participants) | 25 | 23 | 23 | 26 | 22 | 25 | 25 | 24 | 22
  Day 5 | 134.20 (78.692) | 130.30 (58.718) | 112.17 (47.884) | 154.27 (74.707) | 146.41 (76.274) | 128.20 (79.256) | 115.40 (52.401) | 114.25 (61.969) | 121.09 (48.602)
  Day 8: number analyzed (Participants) | 25 | 24 | 24 | 25 | 21 | 25 | 24 | 22 | 23
  Day 8 | 126.44 (123.041) | 124.58 (49.786) | 95.71 (42.796) | 150.40 (76.908) | 128.43 (50.155) | 122.72 (66.459) | 103.50 (48.515) | 130.91 (75.156) | 136.91 (91.378)
  Day 15 | 109.52 (65.672) | 143.96 (70.871) | 123.96 (108.066) | 149.31 (64.392) | 145.91 (79.420) | 125.64 (55.667) | 113.52 (60.601) | 114.25 (54.003) | 130.65 (53.724)
  Day 22: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 22 | 105.56 (45.283) | 119.17 (55.800) | 101.96 (54.725) | 133.65 (48.535) | 144.64 (68.531) | 125.00 (54.636) | 109.04 (49.088) | 113.79 (106.198) | 130.26 (59.246)
  Day 29: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 25 | 25 | 24 | 22
  Day 29 | 97.84 (49.164) | 133.38 (74.370) | 100.04 (39.343) | 147.92 (68.536) | 130.00 (52.743) | 111.24 (46.683) | 142.84 (141.763) | 94.29 (37.698) | 122.09 (49.749)
  Day 36: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 36 | 113.68 (71.769) | 111.25 (45.529) | 96.52 (56.535) | 154.65 (59.929) | 139.95 (79.796) | 115.12 (54.424) | 109.17 (54.052) | 105.67 (38.421) | 158.30 (102.642)
  Day 43 | 108.16 (56.609) | 161.75 (134.409) | 130.71 (124.380) | 159.19 (85.270) | 135.23 (70.762) | 123.80 (52.925) | 119.44 (53.110) | 109.29 (54.365) | 140.61 (73.706)
  Day 50: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Day 50 | 108.12 (65.442) | 126.58 (56.883) | 100.57 (52.553) | 148.50 (77.558) | 121.64 (51.406) | 123.48 (61.199) | 114.22 (53.090) | 113.29 (53.870) | 142.30 (83.014)
  Day 57: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 57 | 94.40 (49.048) | 124.25 (69.357) | 92.52 (45.106) | 139.50 (56.099) | 137.55 (53.502) | 102.28 (33.512) | 117.21 (84.666) | 90.67 (28.925) | 136.78 (67.987)
  Day 71: number analyzed (Participants) | 24 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 71 | 103.13 (51.243) | 125.50 (74.428) | 93.91 (39.340) | 156.27 (65.687) | 139.27 (85.017) | 122.68 (52.192) | 112.13 (56.034) | 103.13 (47.534) | 146.43 (64.368)
  Day 85: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Day 85 | 92.36 (47.872) | 130.25 (78.800) | 95.00 (54.102) | 142.81 (57.891) | 142.45 (60.126) | 118.64 (46.593) | 100.04 (53.185) | 99.92 (40.798) | 119.17 (57.046)
  Day 99: number analyzed (Participants) | 25 | 24 | 22 | 25 | 22 | 25 | 24 | 24 | 23
  Day 99 | 110.56 (57.944) | 128.25 (70.840) | 131.32 (118.340) | 156.84 (70.931) | 137.82 (60.866) | 122.96 (55.697) | 118.17 (63.727) | 115.08 (63.629) | 133.91 (49.879)
  Day 106: number analyzed (Participants) | 25 | 24 | 22 | 25 | 22 | 25 | 23 | 24 | 23
  Day 106 | 97.80 (46.662) | 116.29 (50.480) | 102.59 (50.880) | 131.68 (55.816) | 133.41 (68.902) | 116.16 (55.618) | 109.91 (45.304) | 93.54 (38.520) | 139.00 (53.142)
  Day 113: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 23 | 23
  Day 113 | 101.58 (51.130) | 112.88 (60.824) | 94.39 (34.093) | 141.64 (96.032) | 129.14 (73.031) | 111.72 (53.875) | 116.26 (69.771) | 101.43 (52.274) | 136.61 (64.291)
  Day 127: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 25 | 23 | 24 | 23
  Day 127 | 133.40 (71.046) | 159.25 (101.582) | 115.96 (63.954) | 133.40 (66.304) | 153.14 (62.304) | 138.08 (60.533) | 139.83 (103.182) | 124.50 (86.402) | 159.43 (89.130)
  Day 141: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 24 | 23
  Day 141 | 115.13 (51.964) | 164.79 (129.257) | 123.39 (35.150) | 131.08 (56.266) | 156.27 (76.965) | 135.80 (75.159) | 119.91 (59.343) | 129.13 (70.190) | 137.35 (56.775)
  Day 155: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 23 | 23 | 24 | 23
  Day 155 | 115.44 (39.459) | 164.13 (102.919) | 113.83 (43.209) | 139.44 (65.901) | 149.23 (68.510) | 129.00 (70.010) | 119.91 (61.088) | 133.33 (81.100) | 131.74 (62.736)
  Day 169: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 24 | 23 | 23 | 22
  Day 169 | 120.76 (56.962) | 151.63 (59.252) | 122.43 (65.091) | 149.40 (58.176) | 167.91 (79.436) | 126.67 (60.290) | 166.22 (176.973) | 128.26 (71.260) | 125.41 (36.439)

27. Secondary Outcome: Change From Baseline in Triglyceride (TG) at Day 85 and Day 113
Description: Triglycerides are a type of fat circulating in the blood and account for the majority of the fats circulating in the blood. Fasting was required at least 10 hours before blood sample collection. Baseline was defined as the mean of the last two non-missing measurements collected prior to the first dose of study treatment. Both measurements must be within 10 days prior to the first dose of study treatment; if only one measurement was available 10 days prior to the first dose of study treatment, then that measurement served as the baseline value. Change from baseline = observed value minus baseline value.
Time Frame: Baseline, Day 85, 113
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 26 | 22 | 25 | 25 | 24 | 23
mg/dL
  Change at Day 85: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Change at Day 85 | -28.68 (41.898) | -27.96 (49.754) | -29.52 (40.669) | 2.58 (35.796) | -10.14 (43.129) | -3.76 (37.502) | -15.87 (48.341) | -11.67 (42.519) | -11.22 (23.797)
  Change at Day 113: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 23 | 23
  Change at Day 113 | -20.02 (41.197) | -45.33 (53.285) | -30.13 (48.592) | -0.58 (63.896) | -23.45 (51.443) | -10.68 (27.488) | 0.35 (48.858) | -12.46 (44.128) | 6.22 (32.888)
Statistical Analysis 1: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -35.967, 95% CI 2-sided [-57.463 to -14.472], Standard Error of Mean 10.822
Statistical Analysis 2: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -29.186, 95% CI 2-sided [-51.123 to -7.249], Standard Error of Mean 11.044
Statistical Analysis 3: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -40.010, 95% CI 2-sided [-62.175 to -17.845], Standard Error of Mean 11.160
Statistical Analysis 4: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.614, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 3.170, 95% CI 2-sided [-18.502 to 24.842], Standard Error of Mean 10.906
Statistical Analysis 5: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.221, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -8.563, 95% CI 2-sided [-30.554 to 13.427], Standard Error of Mean 11.067
Statistical Analysis 6: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.303, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -5.649, 95% CI 2-sided [-27.376 to 16.079], Standard Error of Mean 10.933
Statistical Analysis 7: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.067, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -22.003, 95% CI 2-sided [-50.882 to 6.875], Standard Error of Mean 14.530
Statistical Analysis 8: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -41.761, 95% CI 2-sided [-70.934 to -12.588], Standard Error of Mean 14.676
Statistical Analysis 9: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.010, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -34.933, 95% CI 2-sided [-64.410 to -5.456], Standard Error of Mean 14.832
Statistical Analysis 10: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.064, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -17.978, 95% CI 2-sided [-41.282 to 5.326], Standard Error of Mean 11.725
Statistical Analysis 11: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.318, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -5.654, 95% CI 2-sided [-29.311 to 18.004], Standard Error of Mean 11.903
Statistical Analysis 12: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 12]; Test type: Superiority or Other; p = 0.052, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -19.435, 95% CI 2-sided [-42.902 to 4.032], Standard Error of Mean 11.807

28. Secondary Outcome: Percent Change From Baseline in Triglyceride (TG) at Day 85 and Day 113
Description: Triglycerides are a type of fat circulating in the blood and account for the majority of the fats circulating in the blood. Fasting was required at least 10 hours before blood sample collection. Baseline was defined as the mean of the last two non-missing measurements collected prior to the first dose of study treatment. Both measurements must be within 10 days prior to the first dose of study treatment; if only one measurement was available 10 days prior to the first dose of study treatment, then that measurement served as the baseline value. Percent change from baseline = ([observed value divided by baseline value] minus 1) multiplied by 100.
Time Frame: Baseline, Day 85, 113
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 26 | 22 | 25 | 25 | 24 | 23
percent change
  Change at Day 85: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Change at Day 85 | -21.00 (31.109) | -16.85 (28.672) | -23.38 (24.421) | 3.74 (27.803) | -5.20 (23.919) | 2.62 (33.715) | -9.40 (42.868) | -5.21 (35.698) | -9.33 (19.235)
  Change at Day 113: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 23 | 23
  Change at Day 113 | -14.44 (26.916) | -27.65 (26.827) | -17.70 (29.263) | -3.82 (36.247) | -15.23 (24.917) | -8.31 (19.500) | 1.32 (37.694) | -8.47 (35.865) | 4.57 (29.077)
Statistical Analysis 1: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -25.974, 95% CI 2-sided [-41.217 to -10.731], Standard Error of Mean 7.674
Statistical Analysis 2: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -21.110, 95% CI 2-sided [-36.665 to -5.555], Standard Error of Mean 7.831
Statistical Analysis 3: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -31.034, 95% CI 2-sided [-46.758 to -15.310], Standard Error of Mean 7.917
Statistical Analysis 4: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.799, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 8.034, 95% CI 2-sided [-10.948 to 27.015], Standard Error of Mean 9.553
Statistical Analysis 5: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.398, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -2.511, 95% CI 2-sided [-21.748 to 16.727], Standard Error of Mean 9.682
Statistical Analysis 6: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.515, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = 0.369, 95% CI 2-sided [-18.668 to 19.407], Standard Error of Mean 9.580
Statistical Analysis 7: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.128, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -10.056, 95% CI 2-sided [-27.549 to 7.437], Standard Error of Mean 8.801
Statistical Analysis 8: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -24.352, 95% CI 2-sided [-42.008 to -6.695], Standard Error of Mean 8.882
Statistical Analysis 9: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.049, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -14.994, 95% CI 2-sided [-32.858 to 2.870], Standard Error of Mean 8.987
Statistical Analysis 10: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.071, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -13.830, 95% CI 2-sided [-32.368 to 4.709], Standard Error of Mean 9.326
Statistical Analysis 11: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.361, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -3.378, 95% CI 2-sided [-22.191 to 15.435], Standard Error of Mean 9.464
Statistical Analysis 12: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 12]; Test type: Superiority or Other; p = 0.056, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -15.035, 95% CI 2-sided [-33.698 to 3.629], Standard Error of Mean 9.389

29. Secondary Outcome: Non-High Density Lipoprotein- Cholesterol (Non-HDL-C)
Description: Non-HDL-C calculated as total cholesterol minus HDL cholesterol. Fasting was required at least 10 hours before blood sample collection. Baseline was defined as the mean of the last two non-missing measurements collected prior to the first dose of study treatment. Both measurements must be within 10 days prior to the first dose of study treatment; if only one measurement was available 10 days prior to the first dose of study treatment, then that measurement served as the baseline value.
Time Frame: Baseline, Day 5, 8, 15, 22, 29, 36, 43, 50, 57, 71, 85, 99, 106, 113, 127, 141, 155, 169
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 26 | 22 | 25 | 25 | 24 | 23
mg/dL
  Baseline | 159.58 (29.033) | 155.54 (20.706) | 154.71 (22.511) | 163.90 (25.271) | 165.86 (26.655) | 188.72 (30.222) | 182.86 (22.842) | 182.17 (21.217) | 181.17 (23.577)
  Day 5: number analyzed (Participants) | 25 | 23 | 23 | 26 | 22 | 25 | 25 | 24 | 22
  Day 5 | 113.52 (28.259) | 97.78 (25.034) | 98.48 (15.003) | 161.23 (22.059) | 140.77 (26.324) | 154.36 (35.666) | 143.24 (23.520) | 137.50 (28.770) | 189.36 (24.432)
  Day 8: number analyzed (Participants) | 25 | 24 | 24 | 25 | 21 | 25 | 24 | 22 | 23
  Day 8 | 93.24 (22.966) | 79.33 (27.140) | 76.17 (15.222) | 162.16 (29.067) | 131.52 (23.712) | 142.84 (36.478) | 123.25 (25.378) | 122.73 (29.183) | 193.70 (20.424)
  Day 15 | 95.68 (27.248) | 77.88 (27.299) | 57.96 (16.134) | 162.35 (20.558) | 130.27 (19.489) | 138.40 (38.794) | 103.16 (26.742) | 99.13 (22.099) | 191.61 (22.845)
  Day 22: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 22 | 69.92 (23.315) | 58.92 (23.638) | 48.26 (10.037) | 160.04 (19.838) | 130.59 (24.595) | 115.36 (37.861) | 88.71 (24.172) | 88.29 (28.964) | 192.09 (18.757)
  Day 29: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 25 | 25 | 24 | 22
  Day 29 | 81.08 (26.644) | 71.79 (26.662) | 51.09 (14.820) | 159.16 (20.163) | 133.41 (30.589) | 115.52 (38.434) | 90.68 (25.610) | 82.46 (20.659) | 192.59 (23.425)
  Day 36: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 36 | 66.20 (21.848) | 53.38 (22.329) | 44.96 (10.598) | 159.46 (25.221) | 129.32 (29.451) | 103.72 (37.651) | 81.83 (15.898) | 79.42 (26.345) | 184.74 (25.913)
  Day 43 | 79.64 (23.937) | 66.63 (30.685) | 51.46 (14.926) | 157.31 (16.790) | 132.05 (29.005) | 112.60 (37.446) | 88.16 (23.005) | 82.08 (27.547) | 194.30 (22.876)
  Day 50: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Day 50 | 59.92 (17.814) | 52.58 (21.847) | 45.65 (11.276) | 157.62 (22.608) | 130.64 (25.964) | 101.60 (36.427) | 80.30 (20.448) | 78.96 (27.207) | 186.70 (20.220)
  Day 57: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 57 | 75.76 (23.552) | 58.13 (23.709) | 44.26 (9.186) | 153.15 (19.601) | 126.68 (28.919) | 101.80 (35.249) | 86.08 (30.679) | 73.21 (24.568) | 180.17 (17.167)
  Day 71: number analyzed (Participants) | 24 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 71 | 81.83 (28.164) | 58.08 (26.357) | 48.65 (13.110) | 161.54 (22.089) | 134.91 (30.239) | 115.48 (36.001) | 82.25 (22.283) | 76.13 (22.793) | 185.96 (28.798)
  Day 85: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Day 85 | 77.28 (25.268) | 60.04 (23.665) | 49.87 (24.464) | 154.92 (22.289) | 139.05 (36.247) | 110.40 (30.783) | 78.00 (27.144) | 72.17 (18.874) | 175.17 (24.398)
  Day 99: number analyzed (Participants) | 25 | 24 | 22 | 25 | 22 | 25 | 24 | 24 | 23
  Day 99 | 88.56 (28.234) | 66.04 (29.895) | 60.05 (35.754) | 156.36 (18.830) | 133.68 (34.790) | 118.36 (32.875) | 85.29 (30.599) | 74.50 (19.496) | 190.52 (20.551)
  Day 106: number analyzed (Participants) | 25 | 24 | 22 | 25 | 22 | 25 | 23 | 24 | 23
  Day 106 | 64.04 (24.315) | 51.50 (23.178) | 54.14 (28.648) | 154.08 (19.378) | 130.82 (29.301) | 107.76 (31.232) | 77.87 (23.470) | 74.75 (22.115) | 183.35 (19.664)
  Day 113: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 23 | 23
  Day 113 | 82.50 (24.128) | 63.54 (25.086) | 55.78 (27.153) | 146.36 (23.787) | 131.41 (32.515) | 111.80 (30.993) | 83.00 (27.632) | 72.35 (20.232) | 180.65 (16.489)
  Day 127: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 25 | 23 | 24 | 23
  Day 127 | 134.80 (24.100) | 117.42 (37.408) | 85.09 (41.318) | 158.60 (22.504) | 163.36 (33.835) | 164.60 (38.791) | 113.13 (46.332) | 102.75 (33.666) | 191.78 (28.623)
  Day 141: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 24 | 23
  Day 141 | 149.17 (29.556) | 142.08 (32.188) | 119.83 (42.083) | 155.52 (20.490) | 170.41 (37.185) | 187.96 (41.528) | 154.17 (45.140) | 128.96 (44.304) | 191.09 (24.978)
  Day 155: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 23 | 23 | 24 | 23
  Day 155 | 149.60 (26.876) | 144.83 (26.836) | 133.30 (30.526) | 161.80 (21.960) | 169.41 (37.377) | 190.96 (34.453) | 164.83 (34.193) | 144.58 (40.902) | 184.48 (18.030)
  Day 169: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 24 | 23 | 23 | 22
  Day 169 | 155.48 (28.791) | 153.75 (25.535) | 148.52 (27.770) | 159.12 (20.961) | 174.45 (41.877) | 193.88 (33.789) | 183.52 (37.346) | 162.65 (40.341) | 193.59 (17.816)

30. Secondary Outcome: Change From Baseline in Non-High Density Lipoprotein- Cholesterol (Non-HDL-C) at Day 85 and Day 113
Description: Non-HDL-C calculated as total cholesterol minus HDL cholesterol. Fasting was required at least 10 hours before blood sample collection. Baseline was defined as the mean of the last two non-missing measurements collected prior to the first dose of study treatment. Both measurements must be within 10 days prior to the first dose of study treatment; if only one measurement was available 10 days prior to the first dose of study treatment, then that measurement served as the baseline value. Change from baseline = observed value minus baseline value.
Time Frame: Baseline, Day 85, 113
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 26 | 22 | 25 | 25 | 24 | 23
mg/dL
  Change at Day 85: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Change at Day 85 | -82.30 (30.323) | -95.50 (32.345) | -104.07 (27.573) | -8.98 (20.888) | -26.82 (28.796) | -78.32 (33.436) | -104.26 (34.056) | -110.00 (24.274) | -6.00 (24.009)
  Change at Day 113: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 23 | 23
  Change at Day 113 | -77.33 (22.371) | -92.00 (32.099) | -98.15 (28.798) | -18.40 (22.784) | -34.45 (26.242) | -76.92 (35.588) | -99.26 (27.347) | -111.33 (24.646) | -0.52 (20.267)
Statistical Analysis 1: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -76.189, 95% CI 2-sided [-86.975 to -65.403], Standard Error of Mean 5.431
Statistical Analysis 2: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -95.205, 95% CI 2-sided [-106.238 to -84.172], Standard Error of Mean 5.556
Statistical Analysis 3: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -106.077, 95% CI 2-sided [-117.239 to -94.915], Standard Error of Mean 5.622
Statistical Analysis 4: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -71.234, 95% CI 2-sided [-84.390 to -58.077], Standard Error of Mean 6.622
Statistical Analysis 5: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -100.638, 95% CI 2-sided [-113.768 to -87.508], Standard Error of Mean 6.609
Statistical Analysis 6: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -103.386, 95% CI 2-sided [-116.353 to -90.420], Standard Error of Mean 6.525
Statistical Analysis 7: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -61.124, 95% CI 2-sided [-71.813 to -50.435], Standard Error of Mean 5.382
Statistical Analysis 8: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -81.837, 95% CI 2-sided [-92.721 to -70.954], Standard Error of Mean 5.480
Statistical Analysis 9: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -89.683, 95% CI 2-sided [-100.740 to -78.627], Standard Error of Mean 5.567
Statistical Analysis 10: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -76.747, 95% CI 2-sided [-88.902 to -64.593], Standard Error of Mean 6.118
Statistical Analysis 11: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -100.666, 95% CI 2-sided [-112.781 to -88.551], Standard Error of Mean 6.098
Statistical Analysis 12: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 12]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -109.490, 95% CI 2-sided [-121.519 to -97.462], Standard Error of Mean 6.054

31. Secondary Outcome: Percent Change From Baseline in Non-High Density Lipoprotein- Cholesterol (Non-HDL-C) at Day 85 and Day 113
Description: Non-HDL-C calculated as total cholesterol minus HDL cholesterol. Fasting was required at least 10 hours before blood sample collection. Baseline was defined as the mean of the last two non-missing measurements collected prior to the first dose of study treatment. Both measurements must be within 10 days prior to the first dose of study treatment; if only one measurement was available 10 days prior to the first dose of study treatment, then that measurement served as the baseline value. Percent change from baseline = ([observed value divided by baseline value] minus 1) multiplied by 100.
Time Frame: Baseline, Day 85, 113
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 26 | 22 | 25 | 25 | 24 | 23
percent change
  Change at Day 85: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Change at Day 85 | -50.98 (15.662) | -60.62 (17.746) | -67.69 (14.462) | -4.77 (11.716) | -16.20 (16.334) | -41.11 (16.193) | -56.87 (14.745) | -60.17 (10.493) | -2.49 (12.951)
  Change at Day 113: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 23 | 23
  Change at Day 113 | -48.56 (12.284) | -58.57 (17.970) | -63.92 (15.872) | -10.59 (11.977) | -20.67 (15.155) | -40.19 (17.244) | -54.54 (13.671) | -60.43 (11.070) | 0.88 (13.236)
Statistical Analysis 1: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -46.772, 95% CI 2-sided [-53.671 to -39.874], Standard Error of Mean 3.473
Statistical Analysis 2: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -59.200, 95% CI 2-sided [-66.257 to -52.143], Standard Error of Mean 3.554
Statistical Analysis 3: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -66.868, 95% CI 2-sided [-74.007 to -59.730], Standard Error of Mean 3.595
Statistical Analysis 4: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -40.051, 95% CI 2-sided [-47.195 to -32.908], Standard Error of Mean 3.595
Statistical Analysis 5: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -56.009, 95% CI 2-sided [-63.135 to -48.882], Standard Error of Mean 3.587
Statistical Analysis 6: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -57.576, 95% CI 2-sided [-64.618 to -50.533], Standard Error of Mean 3.544
Statistical Analysis 7: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -37.991, 95% CI 2-sided [-44.721 to -31.260], Standard Error of Mean 3.389
Statistical Analysis 8: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -50.856, 95% CI 2-sided [-57.709 to -44.002], Standard Error of Mean 3.451
Statistical Analysis 9: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -56.354, 95% CI 2-sided [-63.315 to -49.393], Standard Error of Mean 3.505
Statistical Analysis 10: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -43.172, 95% CI 2-sided [-50.417 to -35.926], Standard Error of Mean 3.647
Statistical Analysis 11: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -56.698, 95% CI 2-sided [-63.916 to -49.480], Standard Error of Mean 3.633
Statistical Analysis 12: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 12]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -61.305, 95% CI 2-sided [-68.477 to -54.134], Standard Error of Mean 3.609

32. Secondary Outcome: Total Cholesterol (TC) / High Density Lipoprotein- Cholesterol (HDL-C) Ratio
Description: Fasting was required at least 10 hours before blood sample collection. Baseline was defined as the mean of the last two non-missing measurements collected prior to the first dose of study treatment. Both measurements must be within 10 days prior to the first dose of study treatment; if only one measurement was available 10 days prior to the first dose of study treatment, then that measurement served as the baseline value.
Time Frame: Baseline, Day 5, 8, 15, 22, 29, 36, 43, 50, 57, 71, 85, 99, 106, 113, 127, 141, 155, 169
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 26 | 22 | 25 | 25 | 24 | 23
ratio
  Baseline | 4.0118 (0.82813) | 4.0154 (0.92478) | 3.8500 (0.72414) | 3.9629 (0.77435) | 4.0223 (0.81145) | 4.5408 (1.11809) | 4.2558 (1.15512) | 4.2610 (1.08481) | 4.1076 (0.88524)
  Day 5: number analyzed (Participants) | 25 | 23 | 23 | 26 | 22 | 25 | 25 | 24 | 22
  Day 5 | 3.1372 (0.81529) | 2.7861 (0.57451) | 2.7500 (0.38981) | 3.9465 (0.83527) | 3.5668 (0.77085) | 3.9264 (1.11497) | 3.5036 (0.76250) | 3.4029 (0.86267) | 4.3259 (0.99932)
  Day 8: number analyzed (Participants) | 25 | 24 | 24 | 25 | 21 | 25 | 24 | 22 | 23
  Day 8 | 2.7252 (0.63762) | 2.4100 (0.53023) | 2.3083 (0.33483) | 3.8588 (0.92894) | 3.3510 (0.79979) | 3.6024 (1.07004) | 3.1367 (0.80233) | 3.0941 (0.80907) | 4.3374 (0.88617)
  Day 15 | 2.6884 (0.58429) | 2.3754 (0.62550) | 1.9658 (0.33815) | 3.9308 (0.89274) | 3.2700 (0.68229) | 3.4940 (1.02033) | 2.7772 (0.71059) | 2.6050 (0.53948) | 4.3017 (0.84316)
  Day 22: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 22 | 2.2428 (0.53640) | 2.0258 (0.49301) | 1.7730 (0.18504) | 3.8915 (0.75155) | 3.2550 (0.66627) | 3.0676 (0.92151) | 2.4338 (0.43218) | 2.3617 (0.35946) | 4.2822 (0.97569)
  Day 29: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 25 | 25 | 24 | 22
  Day 29 | 2.4020 (0.54386) | 2.2533 (0.64125) | 1.8296 (0.26896) | 3.8852 (0.73498) | 3.3318 (0.70099) | 3.0260 (0.77510) | 2.5780 (0.75738) | 2.2800 (0.37240) | 4.1023 (0.81890)
  Day 36: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 36 | 2.1924 (0.45842) | 1.9300 (0.46830) | 1.7404 (0.18627) | 3.9496 (0.92977) | 3.2882 (0.68375) | 2.8452 (0.78785) | 2.3000 (0.31095) | 2.2529 (0.39114) | 4.2222 (0.97022)
  Day 43 | 2.3688 (0.48338) | 2.1396 (0.61972) | 1.8754 (0.39255) | 3.9338 (0.87409) | 3.3259 (0.70739) | 3.0044 (0.77172) | 2.5124 (0.80082) | 2.3004 (0.42044) | 4.4074 (1.03394)
  Day 50: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Day 50 | 2.0280 (0.36876) | 1.9254 (0.48864) | 1.7443 (0.15406) | 3.9419 (0.98670) | 3.3277 (0.71213) | 2.8300 (0.81738) | 2.2883 (0.38697) | 2.2658 (0.43915) | 4.2909 (0.97014)
  Day 57: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 57 | 2.3148 (0.44657) | 2.0758 (0.63508) | 1.7448 (0.12638) | 3.9596 (0.84943) | 3.2632 (0.60608) | 2.8436 (0.67094) | 2.5708 (1.24941) | 2.2225 (0.37721) | 4.3361 (0.97295)
  Day 71: number analyzed (Participants) | 24 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 71 | 2.3925 (0.57023) | 1.9988 (0.56686) | 1.7709 (0.19489) | 4.0085 (0.93120) | 3.3855 (0.64850) | 3.0528 (0.77095) | 2.3258 (0.34951) | 2.1988 (0.36789) | 4.3791 (1.15180)
  Day 85: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Day 85 | 2.3724 (0.52972) | 2.0721 (0.54913) | 1.8561 (0.49386) | 4.0508 (0.91154) | 3.3986 (0.73940) | 3.1204 (0.72628) | 2.2796 (0.46691) | 2.2142 (0.37394) | 4.2613 (1.08945)
  Day 99: number analyzed (Participants) | 25 | 24 | 22 | 25 | 22 | 25 | 24 | 24 | 23
  Day 99 | 2.4564 (0.54658) | 2.1417 (0.70783) | 2.0305 (0.76914) | 3.7648 (0.83515) | 3.3073 (0.81497) | 3.0868 (0.75654) | 2.4075 (0.70042) | 2.2121 (0.37358) | 4.4200 (1.15874)
  Day 106: number analyzed (Participants) | 25 | 24 | 22 | 25 | 22 | 25 | 23 | 24 | 23
  Day 106 | 2.0476 (0.40004) | 1.8650 (0.50620) | 1.8814 (0.56847) | 3.7912 (0.78337) | 3.2832 (0.72097) | 2.9176 (0.75101) | 2.2517 (0.37291) | 2.1896 (0.37808) | 4.3157 (1.01377)
  Day 113: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 23 | 23
  Day 113 | 2.4688 (0.50001) | 2.1042 (0.55015) | 1.9691 (0.52016) | 3.8248 (0.91875) | 3.2359 (0.65683) | 3.0760 (0.78321) | 2.3639 (0.45213) | 2.2335 (0.42128) | 4.3570 (0.88681)
  Day 127: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 25 | 23 | 24 | 23
  Day 127 | 3.3776 (0.67839) | 3.1533 (0.98795) | 2.4822 (0.91213) | 3.7984 (0.90030) | 3.9132 (0.79683) | 3.9896 (0.99046) | 2.9087 (0.92317) | 2.8208 (1.08222) | 4.4717 (1.06069)
  Day 141: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 24 | 23
  Day 141 | 3.5433 (0.67339) | 3.5242 (0.96281) | 3.0078 (0.91134) | 3.7508 (0.88092) | 3.9841 (0.87530) | 4.4256 (1.20555) | 3.6070 (1.06034) | 3.3500 (1.37776) | 4.2843 (1.17378)
  Day 155: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 23 | 23 | 24 | 23
  Day 155 | 3.6240 (0.63587) | 3.6392 (0.92468) | 3.2748 (0.76307) | 3.9100 (0.92453) | 3.9205 (0.79163) | 4.5057 (1.18175) | 3.8126 (0.99748) | 3.6450 (1.45582) | 4.1804 (1.03516)
  Day 169: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 24 | 23 | 23 | 22
  Day 169 | 3.8140 (0.77275) | 3.7471 (0.82852) | 3.4830 (0.67010) | 3.7436 (0.86236) | 4.0036 (0.99761) | 4.4975 (1.25117) | 4.2000 (1.23292) | 3.8970 (1.40230) | 4.1182 (0.81436)

33. Secondary Outcome: Change From Baseline in Total Cholesterol (TC) / High Density Lipoprotein- Cholesterol (HDL-C) Ratio at Day 85 and Day 113
Description: Fasting was required at least 10 hours before blood sample collection. Baseline was defined as the mean of the last two non-missing measurements collected prior to the first dose of study treatment. Both measurements must be within 10 days prior to the first dose of study treatment; if only one measurement was available 10 days prior to the first dose of study treatment, then that measurement served as the baseline value. Change from baseline = observed value minus baseline value.
Time Frame: Baseline, Day 85, 113
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 26 | 22 | 25 | 25 | 24 | 23
ratio
  Change at Day 85: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Change at Day 85 | -1.6394 (0.69058) | -1.9433 (0.90358) | -1.9835 (0.78766) | 0.0879 (0.43755) | -0.6236 (0.66072) | -1.4204 (0.91892) | -1.8407 (0.85260) | -2.0469 (0.96230) | 0.1537 (0.47755)
  Change at Day 113: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 23 | 23
  Change at Day 113 | -1.5671 (0.65875) | -1.9113 (0.93385) | -1.8704 (0.73630) | -0.1560 (0.53286) | -0.7864 (0.60966) | -1.4648 (0.83864) | -1.7563 (0.74752) | -2.0461 (0.92038) | 0.2493 (0.43772)
Statistical Analysis 1: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -1.69928, 95% CI 2-sided [-1.96175 to -1.43682], Standard Error of Mean 0.13216
Statistical Analysis 2: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -2.07922, 95% CI 2-sided [-2.34622 to -1.81223], Standard Error of Mean 0.13446
Statistical Analysis 3: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Adjusted Mean Difference = -2.23886, 95% CI 2-sided [-2.50795 to -1.96978], Standard Error of Mean 0.13553
Statistical Analysis 4: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -1.43281, 95% CI 2-sided [-1.75689 to -1.10872], Standard Error of Mean 0.16311
Statistical Analysis 5: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -2.01501, 95% CI 2-sided [-2.33718 to -1.69283], Standard Error of Mean 0.16217
Statistical Analysis 6: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -2.11359, 95% CI 2-sided [-2.43230 to -1.79489], Standard Error of Mean 0.16038
Statistical Analysis 7: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -1.35298, 95% CI 2-sided [-1.62324 to -1.08271], Standard Error of Mean 0.13609
Statistical Analysis 8: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -1.79615, 95% CI 2-sided [-2.07001 to -1.52229], Standard Error of Mean 0.13790
Statistical Analysis 9: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -1.86921, 95% CI 2-sided [-2.14575 to -1.59266], Standard Error of Mean 0.13927
Statistical Analysis 10: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -1.57311, 95% CI 2-sided [-1.85788 to -1.28834], Standard Error of Mean 0.14333
Statistical Analysis 11: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -2.00256, 95% CI 2-sided [-2.28521 to -1.71990], Standard Error of Mean 0.14228
Statistical Analysis 12: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 12]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -2.20298, 95% CI 2-sided [-2.48399 to -1.92197], Standard Error of Mean 0.14142

34. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (TC) / High Density Lipoprotein- Cholesterol (HDL-C) Ratio at Day 85 and Day 113
Description: Fasting was required at least 10 hours before blood sample collection. Baseline was defined as the mean of the last two non-missing measurements collected prior to the first dose of study treatment. Both measurements must be within 10 days prior to the first dose of study treatment; if only one measurement was available 10 days prior to the first dose of study treatment, then that measurement served as the baseline value. Percent change from baseline = ([observed value divided by baseline value] minus 1) multiplied by 100.
Time Frame: Baseline, Day 85, 113
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 26 | 22 | 25 | 25 | 24 | 23
percent change
  Change at Day 85: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Change at Day 85 | -39.99 (12.892) | -47.06 (15.152) | -50.43 (13.358) | 2.19 (10.328) | -14.65 (14.740) | -29.51 (16.200) | -43.25 (12.569) | -45.74 (11.961) | 3.81 (10.643)
  Change at Day 113: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 23 | 23
  Change at Day 113 | -38.20 (10.463) | -46.04 (15.705) | -47.68 (13.195) | -3.81 (12.537) | -18.57 (13.541) | -31.07 (14.770) | -41.49 (10.520) | -45.65 (12.114) | 6.98 (12.436)
Statistical Analysis 1: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -41.92915, 95% CI 2-sided [-47.55052 to -36.30778], Standard Error of Mean 2.83037
Statistical Analysis 2: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -51.08604, 95% CI 2-sided [-56.81235 to -45.35973], Standard Error of Mean 2.88356
Statistical Analysis 3: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Adjusted Mean Difference = -55.51600, 95% CI 2-sided [-61.29424 to -49.73777], Standard Error of Mean 2.91014
Statistical Analysis 4: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -33.30375, 95% CI 2-sided [-39.41376 to -27.19373], Standard Error of Mean 3.07498
Statistical Analysis 5: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -47.85210, 95% CI 2-sided [-53.92668 to -41.77751], Standard Error of Mean 3.05746
Statistical Analysis 6: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -48.65686, 95% CI 2-sided [-54.66060 to -42.65313], Standard Error of Mean 3.02097
Statistical Analysis 7: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -33.52920, 95% CI 2-sided [-39.42015 to -27.63826], Standard Error of Mean 2.96599
Statistical Analysis 8: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -43.85680, 95% CI 2-sided [-49.82617 to -37.88744], Standard Error of Mean 3.00531
Statistical Analysis 9: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -46.36865, 95% CI 2-sided [-52.40589 to -40.33142], Standard Error of Mean 3.03981
Statistical Analysis 10: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -38.06019, 95% CI 2-sided [-44.29176 to -31.82863], Standard Error of Mean 3.13610
Statistical Analysis 11: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -48.57807, 95% CI 2-sided [-54.76397 to -42.39217], Standard Error of Mean 3.11350
Statistical Analysis 12: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 12]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -51.87214, 95% CI 2-sided [-58.01968 to -45.72460], Standard Error of Mean 3.09363

35. Secondary Outcome: Apolipoprotein B (ApoB) / Apolipoprotein A-I (ApoA-I) Ratio
Description: as for outcome 32
Time Frame: Baseline, Day 5, 8, 15, 22, 29, 36, 43, 50, 57, 71, 85, 99, 106, 113, 127, 141, 155, 169
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 26 | 22 | 25 | 25 | 24 | 23
ratio
  Baseline | 0.6846 (0.14145) | 0.6606 (0.13665) | 0.6567 (0.12772) | 0.6687 (0.12269) | 0.6775 (0.14076) | 0.7890 (0.17841) | 0.7324 (0.16556) | 0.7167 (0.16058) | 0.6980 (0.13867)
  Day 5: number analyzed (Participants) | 25 | 23 | 23 | 26 | 22 | 25 | 25 | 24 | 22
  Day 5 | 0.4896 (0.14794) | 0.4135 (0.11264) | 0.4222 (0.07116) | 0.6612 (0.12682) | 0.5968 (0.14211) | 0.6428 (0.18885) | 0.5792 (0.11372) | 0.5300 (0.11967) | 0.7100 (0.12642)
  Day 8: number analyzed (Participants) | 25 | 24 | 24 | 25 | 21 | 25 | 24 | 22 | 23
  Day 8 | 0.4044 (0.09862) | 0.3363 (0.11305) | 0.3271 (0.06760) | 0.6660 (0.14947) | 0.5657 (0.14552) | 0.5844 (0.18410) | 0.5017 (0.12310) | 0.4718 (0.13900) | 0.7230 (0.11227)
  Day 15 | 0.4308 (0.12426) | 0.3300 (0.12322) | 0.2450 (0.05649) | 0.6712 (0.13137) | 0.5445 (0.11164) | 0.5776 (0.16885) | 0.4216 (0.11929) | 0.3763 (0.08293) | 0.7226 (0.13404)
  Day 22: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 22 | 0.3136 (0.10610) | 0.2463 (0.09668) | 0.2078 (0.04572) | 0.6773 (0.13012) | 0.5564 (0.13347) | 0.4868 (0.17148) | 0.3629 (0.10897) | 0.3283 (0.09220) | 0.7248 (0.12409)
  Day 29: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 25 | 25 | 24 | 22
  Day 29 | 0.3656 (0.12076) | 0.3058 (0.12721) | 0.2196 (0.05943) | 0.6776 (0.12337) | 0.5609 (0.11924) | 0.4820 (0.14437) | 0.3720 (0.11247) | 0.3254 (0.07524) | 0.7023 (0.11439)
  Day 36: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 36 | 0.2900 (0.09278) | 0.2421 (0.10206) | 0.1983 (0.04376) | 0.6873 (0.15278) | 0.5600 (0.13551) | 0.4428 (0.15255) | 0.3250 (0.06093) | 0.3050 (0.08900) | 0.7048 (0.13413)
  Day 43 | 0.3592 (0.10723) | 0.2800 (0.12399) | 0.2142 (0.05012) | 0.6788 (0.12944) | 0.5805 (0.11978) | 0.4696 (0.15115) | 0.3632 (0.14522) | 0.3188 (0.09124) | 0.7548 (0.16351)
  Day 50: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Day 50 | 0.2668 (0.07669) | 0.2313 (0.10182) | 0.2048 (0.04088) | 0.6804 (0.13489) | 0.5959 (0.13893) | 0.4472 (0.16198) | 0.3283 (0.08917) | 0.3133 (0.09234) | 0.7465 (0.13878)
  Day 57: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 57 | 0.3584 (0.09715) | 0.2642 (0.13319) | 0.2026 (0.04081) | 0.6938 (0.12747) | 0.5682 (0.13297) | 0.4616 (0.15220) | 0.3804 (0.18286) | 0.3196 (0.07765) | 0.7630 (0.13394)
  Day 71: number analyzed (Participants) | 24 | 24 | 23 | 26 | 22 | 25 | 24 | 24 | 23
  Day 71 | 0.3692 (0.12402) | 0.2592 (0.11602) | 0.2157 (0.05281) | 0.6958 (0.13840) | 0.5986 (0.12434) | 0.4976 (0.15592) | 0.3358 (0.07678) | 0.3146 (0.08086) | 0.7500 (0.17328)
  Day 85: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Day 85 | 0.3768 (0.11546) | 0.2696 (0.11705) | 0.2335 (0.10170) | 0.7023 (0.13946) | 0.6132 (0.16069) | 0.5264 (0.14405) | 0.3435 (0.11007) | 0.3125 (0.08125) | 0.7665 (0.18376)
  Day 99: number analyzed (Participants) | 25 | 24 | 22 | 25 | 22 | 25 | 24 | 24 | 23
  Day 99 | 0.3928 (0.12458) | 0.2904 (0.12791) | 0.2491 (0.12432) | 0.6584 (0.13120) | 0.5882 (0.15930) | 0.5164 (0.15168) | 0.3650 (0.15223) | 0.3075 (0.07170) | 0.7883 (0.18622)
  Day 106: number analyzed (Participants) | 25 | 24 | 22 | 25 | 22 | 25 | 23 | 24 | 23
  Day 106 | 0.2908 (0.08450) | 0.2267 (0.10925) | 0.2405 (0.12187) | 0.6716 (0.12925) | 0.5877 (0.15253) | 0.4796 (0.14386) | 0.3322 (0.09130) | 0.3142 (0.08230) | 0.7730 (0.14455)
  Day 113: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 23 | 23
  Day 113 | 0.3888 (0.10343) | 0.2908 (0.11858) | 0.2548 (0.10845) | 0.6556 (0.14192) | 0.5777 (0.12976) | 0.5140 (0.15398) | 0.3557 (0.10710) | 0.3235 (0.08804) | 0.7683 (0.14272)
  Day 127: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 25 | 23 | 24 | 23
  Day 127 | 0.5772 (0.11473) | 0.5029 (0.17571) | 0.3778 (0.19064) | 0.6692 (0.13546) | 0.6950 (0.15732) | 0.7024 (0.18033) | 0.4730 (0.18425) | 0.4325 (0.16469) | 0.7830 (0.15893)
  Day 141: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 24 | 23
  Day 141 | 0.6233 (0.12107) | 0.5938 (0.15786) | 0.5004 (0.19354) | 0.6580 (0.13916) | 0.7082 (0.17595) | 0.7916 (0.20262) | 0.6352 (0.20727) | 0.5375 (0.23022) | 0.7570 (0.17219)
  Day 155: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 23 | 23 | 24 | 23
  Day 155 | 0.6368 (0.11957) | 0.6125 (0.15224) | 0.5574 (0.13288) | 0.6664 (0.13225) | 0.6991 (0.17124) | 0.8148 (0.20102) | 0.6839 (0.19315) | 0.6075 (0.24120) | 0.7452 (0.16318)
  Day 169: number analyzed (Participants) | 25 | 24 | 23 | 25 | 22 | 24 | 23 | 23 | 22
  Day 169 | 0.6640 (0.14350) | 0.6321 (0.14774) | 0.6161 (0.12493) | 0.6424 (0.14621) | 0.6845 (0.17986) | 0.8088 (0.20105) | 0.7178 (0.18178) | 0.6639 (0.22661) | 0.7359 (0.13397)

36. Secondary Outcome: Change From Baseline in Apolipoprotein B (ApoB) / Apolipoprotein A-I (ApoA-I) Ratio at Day 85 and Day 113
Description: as for outcome 33
Time Frame: Baseline, Day 85, 113
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 26 | 22 | 25 | 25 | 24 | 23
ratio
  Change at Day 85: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Change at Day 85 | -0.3078 (0.13144) | -0.3910 (0.15635) | -0.4211 (0.16147) | 0.0337 (0.09054) | -0.0643 (0.11318) | -0.2626 (0.16341) | -0.3748 (0.17224) | -0.4042 (0.14894) | 0.0685 (0.10818)
  Change at Day 113: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 23 | 23
  Change at Day 113 | -0.2998 (0.12105) | -0.3698 (0.16194) | -0.3998 (0.15163) | -0.0170 (0.10303) | -0.0998 (0.09487) | -0.2750 (0.15604) | -0.3626 (0.14553) | -0.3965 (0.15431) | 0.0702 (0.09306)
Statistical Analysis 1: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -0.33157, 95% CI 2-sided [-0.38399 to -0.27916], Standard Error of Mean 0.02639
Statistical Analysis 2: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -0.44402, 95% CI 2-sided [-0.49727 to -0.39077], Standard Error of Mean 0.02682
Statistical Analysis 3: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -0.48314, 95% CI 2-sided [-0.53671 to -0.42956], Standard Error of Mean 0.02698
Statistical Analysis 4: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -0.30542, 95% CI 2-sided [-0.36960 to -0.24124], Standard Error of Mean 0.03230
Statistical Analysis 5: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -0.44143, 95% CI 2-sided [-0.50466 to -0.37821], Standard Error of Mean 0.03183
Statistical Analysis 6: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -0.46235, 95% CI 2-sided [-0.52491 to -0.39980], Standard Error of Mean 0.03148
Statistical Analysis 7: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -0.26949, 95% CI 2-sided [-0.32142 to -0.21755], Standard Error of Mean 0.02615
Statistical Analysis 8: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -0.37493, 95% CI 2-sided [-0.42754 to -0.32231], Standard Error of Mean 0.02649
Statistical Analysis 9: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -0.41199, 95% CI 2-sided [-0.46512 to -0.35886], Standard Error of Mean 0.02676
Statistical Analysis 10: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -0.31806, 95% CI 2-sided [-0.37723 to -0.25888], Standard Error of Mean 0.02979
Statistical Analysis 11: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -0.42583, 95% CI 2-sided [-0.48409 to -0.36758], Standard Error of Mean 0.02932
Statistical Analysis 12: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -0.45501, 95% CI 2-sided [-0.51287 to -0.39715], Standard Error of Mean 0.02912

37. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B (ApoB) / Apolipoprotein A-I (ApoA-I) Ratio at Day 85 and Day 113
Description: as for outcome 34
Time Frame: Baseline, Day 85, 113
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 26 | 22 | 25 | 25 | 24 | 23
percent change
  Change at Day 85: number analyzed (Participants) | 25 | 24 | 23 | 26 | 22 | 25 | 23 | 24 | 23
  Change at Day 85 | -44.37 (16.358) | -58.47 (19.271) | -63.09 (16.240) | 5.51 (12.823) | -9.13 (16.695) | -32.09 (18.463) | -50.97 (16.380) | -55.16 (11.927) | 10.41 (15.319)
  Change at Day 113: number analyzed (Participants) | 24 | 24 | 23 | 25 | 22 | 25 | 23 | 23 | 23
  Change at Day 113 | -43.21 (13.147) | -55.05 (19.756) | -60.32 (15.924) | -2.03 (14.326) | -14.00 (14.205) | -34.11 (18.505) | -49.84 (13.744) | -53.65 (13.386) | 11.47 (16.250)
Statistical Analysis 1: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -49.42411, 95% CI 2-sided [-56.83019 to -42.01803], Standard Error of Mean 3.72907
Statistical Analysis 2: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -66.63383, 95% CI 2-sided [-74.16086 to -59.10681], Standard Error of Mean 3.79050
Statistical Analysis 3: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Adjusted Mean Difference = -71.72901, 95% CI 2-sided [-79.30431 to -64.15371], Standard Error of Mean 3.81541
Statistical Analysis 4: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -43.56596, 95% CI 2-sided [-51.35899 to -35.77293], Standard Error of Mean 3.92236
Statistical Analysis 5: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -62.34926, 95% CI 2-sided [-70.02607 to -54.67245], Standard Error of Mean 3.86432
Statistical Analysis 6: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -65.06617, 95% CI 2-sided [-72.65818 to -57.47415], Standard Error of Mean 3.82052
Statistical Analysis 7: Comparison: Atorvastatin + PF-04950615 50 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -40.52435, 95% CI 2-sided [-47.81299 to -33.23571], Standard Error of Mean 3.66973
Statistical Analysis 8: Comparison: Atorvastatin + PF-04950615 100 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -56.14495, 95% CI 2-sided [-63.52668 to -48.76322], Standard Error of Mean 3.71641
Statistical Analysis 9: Comparison: Atorvastatin + PF-04950615 150 mg vs Atorvastatin + PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -61.56370, 95% CI 2-sided [-69.02510 to -54.10230], Standard Error of Mean 3.75690
Statistical Analysis 10: Comparison: PF-04950615 50 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -46.34109, 95% CI 2-sided [-54.61427 to -38.06792], Standard Error of Mean 4.16385
Statistical Analysis 11: Comparison: PF-04950615 100 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -61.37890, 95% CI 2-sided [-69.52338 to -53.23443], Standard Error of Mean 4.09957
Statistical Analysis 12: Comparison: PF-04950615 150 mg vs PF-04950615 Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; One-sided p-values (unadjusted for multiplicity) was derived from the MMRM model; Adjusted Mean Difference = -64.67274, 95% CI 2-sided [-72.75728 to -56.58820], Standard Error of Mean 4.06866

38. Secondary Outcome: Percentage of Participants Achieving Low-density Lipoprotein Cholesterol (LDL-C) Less Than (<) 10, 25, 40, 70 and 100 Milligram Per Deciliter
Description: LDL-C is cholesterol in the bloodstream that is carried by low density lipoprotein. Fasting was required at least 10 hours before blood sample collection.
Time Frame: Baseline up to Day 113
Population: FAS included all the participants who were randomized and administered at least 1 dose of study treatment. The outcome measure was planned to be analyzed for all the reporting groups except Atorvastatin + Ezetimibe 10 mg.
Measure: Number; unit: percentage of participants
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 26 | 25 | 25 | 24 | 23
percentage of participants
  LDL-C <10 mg/dL | 0.0 | 4.2 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  LDL-C <25 mg/dL | 12.0 | 66.7 | 58.3 | 0.0 | 0.0 | 0.0 | 20.8 | 0.0
  LDL-C <40 mg/dL | 84.0 | 91.7 | 95.8 | 0.0 | 12.0 | 36.0 | 41.7 | 0.0
  LDL-C <70 mg/dL | 96.0 | 100.0 | 100.0 | 0.0 | 64.0 | 92.0 | 87.5 | 0.0
  LDL-C <100 mg/dL | 100.0 | 100.0 | 100.0 | 23.1 | 92.0 | 100.0 | 100.0 | 4.3

39. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) or Serious Adverse Events (SAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. TEAEs are events between first dose of study drug and up to Day 169 that were absent before treatment or that worsened relative to pretreatment state. Adverse events included treatment emergent injection site adverse events and any clinically significant abnormal laboratory value.
Time Frame: Baseline up to Day 169
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 26 | 22 | 25 | 25 | 24 | 23
participants
  AEs | 17 | 16 | 13 | 13 | 5 | 16 | 16 | 15 | 11
  SAEs | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0

40. Secondary Outcome: Number of Participants With Anti-Drug Antibody (ADA) Response
Description: Participants tested positive for ADA response on at least one post-baseline visit were reported. Participants with ADA titer level >=6.23 for PF-04950615 were considered ADA positive.
Time Frame: Baseline up to Day 169
Population: Safety analysis set included all randomized and non-randomized participants who were administered at least 1 dose of study treatment. This outcome measure was planned to be analyzed for all the reporting groups except for Atorvastatin + Ezetimibe 10 mg.
Measure: Number; unit: participants
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 0 | 25 | 25 | 24 | 0
participants | 14 | 6 | 14 |  | 13 | 16 | 11 |

41. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of PF-04950615
Description: Area under the plasma concentration time-curve from time zero to end of dosing interval (tau). This outcome measure was to be analyzed in participants who received at least 1 dose of the PF-04950615.
Time Frame: Single dose (Day 1: pre-dose, 24, 48, 72, 96, 120, 144, 168 hour (hr) post-dose), Multiple dose (Day 99: pre-dose, 24, 72, 120, 168, 336, 504, 672, 1008 hr post-dose)
Population: The pharmacokinetic (PK) parameter analysis population included participants with full PK sampling in FAS who had at least 1 of the PF-04950615 PK parameters of interest. Here, 'Number analyzed' = Participants evaluable for this outcome measure at specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*day per milliliter(mcg*day/mL)
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg
Number analyzed (Participants) | 12 | 12 | 13 | 11 | 12 | 12
microgram*day per milliliter(mcg*day/mL)
  Single dose | 32.98 (57) | 52.33 (49) | 77.11 (43) | 32.97 (42) | 51.49 (46) | 82.05 (45)
  Multiple dose: number analyzed (Participants) | 10 | 8 | 8 | 10 | 11 | 12
  Multiple dose | 63.54 (40) | 92.46 (127) | 242.5 (81) | 63.74 (57) | 136.6 (32) | 273.5 (100)

42. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] of PF-04950615
Description: Area under the plasma concentration-time profile from time zero extrapolated to infinite time. This outcome measure was to be analyzed in participants who received at least 1 dose of the PF-04950615.
Time Frame: Multiple dose (Day 99: pre-dose, 24, 72, 120, 168, 336, 504, 672, 1008 hr post-dose)
Population: The PK parameter analysis population included participants with full PK sampling in FAS who had at least 1 of the PF-04950615 PK parameters of interest. Here, number of participants analyzed (N) signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*day/mL
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg
Number analyzed (Participants) | 10 | 7 | 8 | 9 | 11 | 7
mcg*day/mL | 94.83 (46) | 176.9 (144) | 469.5 (90) | 111.7 (63) | 237.4 (41) | 248.4 (76)

43. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of PF-04950615
Description: Area under the plasma concentration-time profile from time zero to the time of the last quantifiable concentration. This outcome measure was to be analyzed in participants who received at least 1 dose of the PF-04950615.
Time Frame: Multiple dose (Day 99: pre-dose, 24, 72, 120, 168, 336, 504, 672, 1008 hr post-dose)
Population: The PK parameter analysis population included participants with full PK sampling in FAS who had at least 1 of the PF-04950615 PK parameters of interest. Here, N signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*day/mL
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg
Number analyzed (Participants) | 10 | 8 | 8 | 10 | 11 | 12
mcg*day/mL | 87.86 (49) | 140.3 (145) | 434.2 (91) | 96.32 (65) | 220.9 (39) | 486.7 (143)

44. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-04950615
Description: This outcome measure was to be analyzed in participants who received at least 1 dose of the PF-04950615.
Time Frame: Single dose (Day 1: pre-dose, 24, 48, 72, 96, 120, 144, 168 hr post-dose), Multiple dose (Day 99: pre-dose, 24, 72, 120, 168, 336, 504, 672, 1008 hr post-dose)
Population: The PK parameter analysis population included participants with full PK sampling in FAS who had at least 1 of the PF-04950615 PK parameters of interest. Here, 'Number analyzed' = Participants evaluable for this outcome measure at specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (mcg/mL)
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg
Number analyzed (Participants) | 12 | 12 | 13 | 11 | 12 | 12
microgram per milliliter (mcg/mL)
  Single dose | 3.173 (61) | 5.074 (50) | 7.382 (45) | 2.994 (44) | 4.744 (47) | 7.726 (42)
  Multiple dose: number analyzed (Participants) | 10 | 8 | 8 | 10 | 11 | 12
  Multiple dose | 6.197 (36) | 8.343 (119) | 21.91 (76) | 5.874 (55) | 12.22 (29) | 23.64 (88)

45. Secondary Outcome: Minimum Observed Plasma Trough Concentration (Cmin) of PF-04950615
Description: This outcome measure was to be analyzed in participants who received at least 1 dose of the PF-04950615.
Time Frame: Multiple dose (Day 99: pre-dose, 24, 72, 120, 168, 336, 504, 672, 1008 hr post-dose)
Population: as for outcome 43
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg
Number analyzed (Participants) | 10 | 8 | 8 | 10 | 11 | 12
mcg/mL | 2.176 (65) | 4.041 (147) | 12.95 (94) | 2.858 (64) | 6.571 (40) | 13.47 (139)

46. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-04950615
Description: This outcome measure was to be analyzed in participants who received at least 1 dose of the PF-04950615.
Time Frame: as for outcome 41
Population: as for outcome 44
Measure: Median (Full Range); unit: day
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg
Number analyzed (Participants) | 12 | 12 | 13 | 11 | 12 | 12
day
  Single dose | 4.01 [3.00 to 5.96] | 4.97 [3.94 to 7.00] | 5.94 [1.94 to 7.00] | 5.94 [3.94 to 6.95] | 5.45 [2.95 to 6.94] | 6.94 [2.96 to 14.0]
  Multiple dose: number analyzed (Participants) | 10 | 8 | 8 | 10 | 11 | 12
  Multiple dose | 3.03 [2.92 to 6.98] | 2.98 [1.00 to 4.97] | 2.97 [0.964 to 4.99] | 2.99 [0.985 to 7.06] | 2.98 [0.988 to 4.98] | 4.98 [2.97 to 7.00]

47. Secondary Outcome: Terminal Elimination Half-Life (t1/2) of PF-04950615
Description: Terminal elimination half-life is the time measured for the plasma concentration to decrease by one half. This outcome measure was to be analyzed in participants who received at least 1 dose of the PF-04950615.
Time Frame: Multiple dose (Day 99: pre-dose, 24, 72, 120, 168, 336, 504, 672, 1008 hr post-dose)
Population: as for outcome 43
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg
Number analyzed (Participants) | 10 | 7 | 8 | 9 | 11 | 7
day | 7.716 (1.7594) | 9.471 (2.2889) | 10.56 (1.5934) | 9.404 (2.1454) | 9.570 (2.2338) | 9.333 (2.7535)

48. Secondary Outcome: Plasma Concentration of Proprotein Convertase Subtilisin/Kexin Type 9 (PCSK9)
Description: Concentration versus time summary was calculated by setting concentration values below the lower limit of quantification (LLQ =6.99 nanogram per milliliter [ng/mL]) to zero. Summary statistics were not to be presented if number of observations above lower limit of quantification (NALQ) =0. Here, 'Number analyzed' = Participants evaluable for this outcome measure at specified time points.
Time Frame: Day 1, 5, 8, 15, 22, 29, 36, 43, 50, 57, 71, 85, 99, 106, 113, 127, 141
Population: PK concentration population included participants in FAS who have at least 1 concentration of either PF-04950615, PCSK9 or atorvastatin or its active metabolites. This outcome measure was planned to be analyzed for all the reporting groups except for Atorvastatin + Ezetimibe 10 mg.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Number analyzed (Participants) | 25 | 24 | 24 | 26 | 25 | 25 | 24 | 23
ng/mL
  Day 1: number analyzed (Participants) | 25 | 24 | 24 | 26 | 25 | 24 | 24 | 23
  Day 1 | 266.64 (61.5494) | 261.23 (72.3625) | 285.96 (75.7940) | 269.19 (66.8377) | 228.80 (49.9983) | 215.50 (43.0086) | 234.42 (77.5410) | 210.22 (48.5536)
  Day 5: number analyzed (Participants) | 25 | 23 | 23 | 26 | 25 | 25 | 24 | 22
  Day 5 | 2292.2 (676.414) | 2152.6 (451.749) | 1997.7 (563.722) | 291.77 (65.8011) | 1952.5 (527.661) | 1775.4 (531.225) | 1712.0 (458.574) | 240.41 (63.093)
  Day 8: number analyzed (Participants) | 25 | 24 | 24 | 26 | 25 | 23 | 23 | 23
  Day 8 | 2711.2 (614.649) | 2701.9 (568.958) | 2539.5 (587.196) | 292.19 (62.5108) | 2490.4 (573.777) | 2297.7 (521.003) | 2306.7 (594.409) | 240.22 (53.5842)
  Day 15: number analyzed (Participants) | 25 | 24 | 24 | 26 | 25 | 23 | 23 | 23
  Day 15 | 2539.8 (558.369) | 3198.1 (897.565) | 3291.9 (624.935) | 303.42 (47.9418) | 2590.6 (601.052) | 3030.8 (715.193) | 2966.7 (713.934) | 224.43 (57.6903)
  Day 22: number analyzed (Participants) | 20 | 22 | 20 | 25 | 16 | 21 | 21 | 17
  Day 22 | 3451.7 (872.597) | 3297.3 (701.137) | 3166.5 (663.295) | 295 (71.6996) | 3117.4 (582.258) | 2971.6 (669.215) | 2726.7 (616.409) | 218.82 (41.2647)
  Day 29: number analyzed (Participants) | 25 | 23 | 22 | 25 | 24 | 23 | 24 | 23
  Day 29 | 2844.2 (684.693) | 3224.8 (868.760) | 3419.8 (715.001) | 275 (57.6888) | 3050.0 (534.176) | 3095.5 (647.481) | 2955.6 (678.703) | 230.09 (44.1742)
  Day 36: number analyzed (Participants) | 20 | 20 | 21 | 24 | 23 | 22 | 23 | 22
  Day 36 | 3446.2 (825.704) | 3310.7 (732.706) | 3248.5 (660.213) | 304.75 (48.529) | 3237.0 (694.727) | 3011.2 (578.469) | 2761.4 (601.567) | 233.09 (56.7693)
  Day 43: number analyzed (Participants) | 25 | 23 | 22 | 26 | 24 | 23 | 24 | 23
  Day 43 | 2900.9 (653.572) | 3406.3 (765.437) | 3391.9 (717.922) | 303.54 (81.0823) | 3278.9 (693.207) | 3302.5 (584.658) | 3016.9 (772.615) | 239.13 (43.8782)
  Day 50: number analyzed (Participants) | 22 | 22 | 19 | 24 | 22 | 22 | 21 | 20
  Day 50 | 3394.8 (750.557) | 3297.2 (654.384) | 3230.9 (716.416) | 293.38 (66.9138) | 3148.5 (541.230) | 3001.3 (696.256) | 2820.3 (693.130) | 237.40 (68.2421)
  Day 57: number analyzed (Participants) | 25 | 23 | 21 | 26 | 23 | 22 | 24 | 23
  Day 57 | 2779.2 (698.727) | 3204.8 (699.490) | 3390.6 (1149.17) | 277.69 (70.6132) | 2910.6 (531.493) | 3026.4 (708.490) | 2791.9 (633.717) | 220.13 (66.99)
  Day 71: number analyzed (Participants) | 24 | 23 | 21 | 26 | 23 | 22 | 24 | 23
  Day 71 | 2889.6 (542.831) | 3241.2 (724.363) | 3280.5 (727.932) | 285.81 (45.5315) | 3066.8 (693.445) | 3197.1 (575.162) | 2887.6 (684.734) | 355.17 (556.079)
  Day 85: number analyzed (Participants) | 25 | 23 | 21 | 26 | 23 | 22 | 24 | 23
  Day 85 | 2727.0 (635.595) | 3166.3 (736.216) | 3198.9 (827.313) | 276.31 (72.3396) | 2898.7 (551.114) | 2934.1 (548.311) | 2787.9 (812.792) | 269.61 (201.161)
  Day 99: number analyzed (Participants) | 24 | 16 | 13 | 25 | 23 | 22 | 23 | 23
  Day 99 | 2915.1 (711.932) | 3242.9 (684.758) | 3259.6 (754.730) | 326.08 (78.8759) | 3119.2 (665.408) | 3149.3 (590.228) | 2918.9 (752.647) | 252.13 (72.1011)
  Day 106: number analyzed (Participants) | 24 | 15 | 12 | 24 | 23 | 23 | 21 | 22
  Day 106 | 3326.7 (611.790) | 3138.9 (604.177) | 2864.0 (596.757) | 283.67 (58.9079) | 3165.7 (786.665) | 2755.7 (549.755) | 2566.5 (483.133) | 242.23 (59.4266)
  Day 113: number analyzed (Participants) | 22 | 15 | 12 | 24 | 23 | 23 | 19 | 22
  Day 113 | 2727.3 (710.746) | 2919.0 (511.959) | 2910.3 (609.380) | 267.71 (68.1498) | 2908.4 (639.771) | 3009.8 (685.462) | 2683.9 (574.842) | 222.05 (46.0574)
  Day 127: number analyzed (Participants) | 24 | 15 | 12 | 25 | 23 | 23 | 21 | 23
  Day 127 | 1429.8 (599.406) | 2148.7 (1062.32) | 3030.7 (607.610) | 281.40 (95.7562) | 1778.9 (872.368) | 2556.0 (772.015) | 2769.7 (736.453) | 249.87 (63.2113)
  Day 141: number analyzed (Participants) | 24 | 15 | 13 | 25 | 23 | 23 | 21 | 23
  Day 141 | 736.63 (297.087) | 1382.8 (892.457) | 2851.0 (1373.69) | 290.16 (84.2168) | 1056.5 (545.337) | 1477.0 (816.342) | 2368.7 (1106.62) | 20.043 (68.7012)

ADVERSE EVENTS:
Groups:
- Atorvastatin + Ezetimibe 10 mg QD PO: Participants received Atorvastatin plus Ezetimibe 10 mg oral administration once daily for 16 week (open).
Arm/Group | Atorvastatin + PF-04950615 50 mg | Atorvastatin + PF-04950615 100 mg | Atorvastatin + PF-04950615 150 mg | Atorvastatin + PF-04950615 Placebo | Atorvastatin + Ezetimibe 10 mg QD PO | PF-04950615 50 mg | PF-04950615 100 mg | PF-04950615 150 mg | PF-04950615 Placebo
Serious Adverse Events (participants affected / at risk) | 1/25 | 0/24 | 0/24 | 1/26 | 0/22 | 0/25 | 1/25 | 0/24 | 0/23
Other Adverse Events (participants affected / at risk) | 10/25 | 12/24 | 12/24 | 10/26 | 2/22 | 11/25 | 11/25 | 11/24 | 9/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atorvastatin + PF-04950615 50 mg (N=25) | Atorvastatin + PF-04950615 100 mg (N=24) | Atorvastatin + PF-04950615 150 mg (N=24) | Atorvastatin + PF-04950615 Placebo (N=26) | Atorvastatin + Ezetimibe 10 mg QD PO (N=22) | PF-04950615 50 mg (N=25) | PF-04950615 100 mg (N=25) | PF-04950615 150 mg (N=24) | PF-04950615 Placebo (N=23)
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Atorvastatin + PF-04950615 50 mg (N=25) | Atorvastatin + PF-04950615 100 mg (N=24) | Atorvastatin + PF-04950615 150 mg (N=24) | Atorvastatin + PF-04950615 Placebo (N=26) | Atorvastatin + Ezetimibe 10 mg QD PO (N=22) | PF-04950615 50 mg (N=25) | PF-04950615 100 mg (N=25) | PF-04950615 150 mg (N=24) | PF-04950615 Placebo (N=23)
Injection site erythema (General disorders) | 2 | 6 | 8 | 0 | 0 | 4 | 7 | 6 | 1
Injection site haemorrhage (General disorders) | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 0
Injection site pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Injection site pruritus (General disorders) | 2 | 4 | 7 | 0 | 0 | 4 | 6 | 5 | 0
Injection site swelling (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 5 | 1 | 1 | 5 | 1 | 3 | 4 | 2 | 4
Pharyngitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 5 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 0 | 0 | 3 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0 | 3 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ejaculation disorder (Reproductive system and breast disorders) | 0/17 | 0/14 | 1/12 | 0/13 | 0/12 | 0/10 | 0/15 | 0/13 | 0/18 — Gender specific adverse event.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.